CLINICAL TRIAL: NCT01975389
Title: Phase 3 Multi Center, Double Blind, Randomized, Placebo Controlled, Parallel Group Evaluation Of The Efficacy, Safety, And Tolerability Of Bococizumab (Pf-04950615), In Reducing The Occurrence Of Major Cardiovascular Events In High Risk Subjects
Brief Title: The Evaluation of Bococizumab (PF-04950615; RN316) in Reducing the Occurrence of Major Cardiovascular Events in High Risk Subjects
Acronym: SPIRE-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1481038; CV OUTCOMES 2; 2013-002795-41 (EudraCT Number)
Record Dates: First submitted 2013-10-21; First posted 2013-11-04 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Disease
Keywords: myocardial infarction; stroke; hyperlipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; Hyperlipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- bococizumab (PF-04950615) (Experimental): 150 mg, every 2 weeks, subcutaneous.
  Interventions: Drug: bococizumab (PF-04950615)
- Placebo (Placebo Comparator): Placebo comparator, every 2 weeks, subcutaneous.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bococizumab (PF-04950615) — 150 mg, every 2 weeks, subcutaneous. The duration of the treatment period will depend upon reaching the targeted number of adjudicated and confirmed CV outcome events, approximately 3 to 4 years after the entry of first subject into the study.
  Other Names: RN316
  Arms: bococizumab (PF-04950615)
Drug: Placebo — Placebo comparator, every 2 weeks, subcutaneous. The duration of the treatment period will depend upon reaching the targeted number of adjudicated and confirmed CV outcome events, approximately 3 to 4 years after the entry of first subject into the study.
  Arms: Placebo

SUMMARY:
This study evaluates the PCSK9 inhibitor, Bococizumab (PF-04950615;RN316), compared to placebo, in reducing the occurrrence of major cardiovascular events, including cardiovascular death, myocardial infarction, stroke, and unstable angina requiring urgent revascularization in high risk subjects who are receiving background lipid lowering therapy and have cholesterol laboratory values of LDL-C >/= 100 mg/dL (2.6 mmol/L) or non-HDL-C >/=130 mg/dL (3.4 mmol/L).

DETAILED DESCRIPTION:
The trial was terminated prematurely on November 1, 2016, due to the emerging clinical profile and the evolving treatment and market landscape for lipid-lowering agents. These indicated that bococizumab was not likely to provide value to patients, physicians, or shareholders. The decision was not based on a recommendation by the independent Data Monitoring Committee to stop the program.

ELIGIBILITY:
Inclusion Criteria:

* Must be on background lipid lowering treatment.
* Must be at high risk of a CV event.
* Must have an LDL C >/=100 mg/dL (2.6 mmol/L) OR non HDL C >/=130 mg/dL (3.4 mmol/L).

Exclusion Criteria:

* Planned coronary (PCI or CABG) or other arterial revascularization.
* New York Heart Association Class IV congestive heart failure or left ventricular ejection fraction < 25% by cardiac imaging.
* Chronic renal insufficiency with creatinine clearance of <30 ml/min/1.73m^2 by MDRD formula or with end state renal disease on dialysis.
* History of hemorrhagic stroke.
* Prior exposure to bococizumab or other investigational PCSK9 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10564 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1587):
- United States (515):
  - Ernest Hendrix, MD, PC, Athens, Alabama
  - North Alabama Research Center, LLC, Athens, Alabama
  - Central Alabama Research, Birmingham, Alabama
  - Clinical Research Advantage, Inc./Simon Williamson Clinic, Birmingham, Alabama
  - The Kirklin Clinic, Birmingham, Alabama
  - Birmingham Heart Clinic, P.C., Birmingham, Alabama
  - University of Alabama at Birmingham (Drug Shipment), Birmingham, Alabama
  - Appalachian Cardiovascular Associates, Fort Payne, Alabama
  - Fundamental Research, LLC, Gulf Shores, Alabama
  - Avant Research Associates, LLC, Guntersville, Alabama
  - Boyett Health Services, Hamilton, Alabama
  - The Office of Saadat Ansari MD LLC, Huntsville, Alabama
  - CB Flock Research Corporation, Mobile, Alabama
  - Alaska Heart Institute, Anchorage, Alaska
  - Phoenix Heart, PLLC, Glendale, Arizona
  - Arrowhead Internal Medicine, Glendale, Arizona
  - Clinical Research Advantage, Inc./Family Practice Specialists, Ltd., Phoenix, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Clinical Research Advantage, Inc. (Administrative Mailing Only), Tempe, Arizona
  - Southwest Heart Group, Tucson, Arizona
  - Arizona Endocrine and Rheumatology Associates, Tucson, Arizona
  - Arkansas Heart Hospital Clinic, Little Rock, Arkansas
  - Arkansas Site Management Services, LLC, Little Rock, Arkansas
  - Cardiology Consultants of Orange County Medical Group, Inc., Anaheim, California
  - Premier Valley Medical Group, Bakersfield, California
  - Cardiovascular Research Foundation of Southern California, Beverly Hills, California
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - Southbay Pharma Research, Buena Park, California
  - Pioneer Medical Group, Cerritos, California
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Atlantic Ave Medical Clinic Inc., Cudahy, California
  - Multani Medical Group, Downey, California
  - Triwest Research Associates, LLC, El Cajon, California
  - Diagnamics Inc., Encinitas, California
  - T. Joseph Raoof, Md, Inc/Encino Research Center, Encino, California
  - Aviva Research, Escondido, California
  - Valley Research, Fresno, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - Omnibus Clinical Research, La Palma, California
  - Alliance Research Centers, Laguna Hills, California
  - Prime Care Clinical Research Center, Laguna Hills, California
  - Clinical Trials Research, Lincoln, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - American Institute of Research, Los Angeles, California
  - Intermed Group, Los Angeles, California
  - Academic Medical Research Institute, Los Angeles, California
  - Eastside Clinical Research Associates, Los Angeles, California
  - Richard S. Cherlin, MD, Los Gatos, California
  - Facey Medical Foundation, Mission Hills, California
  - California Medical Research Associates Inc., Northridge, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Diabetes Associates Medical Group, Orange, California
  - Saviers Medical Group, Port Hueneme, California
  - California Research Foundation, San Diego, California
  - San Diego Family Care dba Linda Vista Health Center, San Diego, California
  - San Diego Family Care, San Diego, California
  - Ritchken & First Md's, San Diego, California
  - Wetlin Research Associates, Inc., San Diego, California
  - West Coast Research LLC, San Ramon, California
  - Syrentis Clinical Research, Santa Ana, California
  - Coastal Biomedical Research, Inc., Santa Monica, California
  - Encompass Clinical Research, Spring Valley, California
  - St. Joseph's Medical Associates, Stockton, California
  - Westlake Medical Research, Thousand Oaks, California
  - Harbor-UCLA Medical Center - Torrance, Torrance, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Bayview Research Group, Valley Village, California
  - Coastal Metabolic Research Centre, Ventura, California
  - Ventura Clinical Trials, Ventura, California
  - Clinical Research Advantage, Inc. / Cassidy Medical Group - Vista, Vista, California
  - Allianz Research Institute, Westminster, California
  - American Institute of Research Studies, Whittier, California
  - American Institute of Research, Whittier, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Elite Clinical Trials, Incorporated, Wildomar, California
  - Colorado Springs Health Partners, Colorado Springs, Colorado
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Memorial Hospital: University of Colorado Health, Colorado Springs, Colorado
  - Lynn Institute of Denver, Denver, Colorado
  - Western Colorado Research, LLC, Glenwood Springs, Colorado
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Connecticut Clinical Research, LLC, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Cardiology Associates of Fairfield County, PC, Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Alfieri Cardiology, Wilmington, Delaware
  - ACRC - Cardiology, Atlantis, Florida
  - GulfCoast Endocrine and Diabetes Center, Clearwater, Florida
  - Morton Plant Mease Health Care, Inc. Cardiovascular Research, Clearwater, Florida
  - Team Medical Research, Coral Gables, Florida
  - The Heart Group, PA, Daytona Beach, Florida
  - Cardiology Associates Research Company, Daytona Beach, Florida
  - The Cardiology Center, Delray Beach, Florida
  - Continental Research Corp, Doral, Florida
  - Care Research Center Inc, Doral, Florida
  - Integrity Clinical Research, LLC, Doral, Florida
  - Moonshine Research Center, Inc., Doral, Florida
  - Invesclinic, LLC, Fort Lauderdale, Florida
  - The Office of Dr. Alan Graff, MD, PA, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - The Office of Maxine E. Hamilton, MD, PA, Fort Lauderdale, Florida
  - State Of The Art Research, LLC, Hialeah, Florida
  - Direct Helpers Medical Center Inc, Hialeah, Florida
  - Research Physicians Network Alliance, Hollywood, Florida
  - Pines Clinical Research, Inc., Hollywood, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - River City Clinical Research, Jacksonville, Florida
  - East Coast Institute for Reserach, LLC, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - The Office of Rachel Day, Jacksonville, Florida
  - Baker-Gilmore Cardiovascular Institute, Jacksonville, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - The Heart Institute at Largo, Largo, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Future Clinical Research, Inc., Miami, Florida
  - Advanced Clinical Research of Miami (ACROM) International, Miami, Florida
  - Project4Research, Inc, Miami, Florida
  - A & L Clinical Research, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Team Medical Research, Inc., Miami, Florida
  - Team Medical Research, Miami, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Florida Medical Center & Research, Inc., Miami, Florida
  - Medical Research Center, Miami, Florida
  - Nuren Medical & Research Center, Miami, Florida
  - Doctors Research Institute, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Coast Research Institute, Miami, Florida
  - My Community Research Center, Inc., Miami, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Research Institute of South Florida, Inc., Miami, Florida
  - A & O Research Center, Inc., Miami, Florida
  - BWell Research Center, Miami, Florida
  - Pharmacology International Research, Inc., Miami, Florida
  - Advanced Clinical Research, Miami, Florida
  - South Florida Research Group, LLC, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Kendall South Medical Center, Inc, Miami, Florida
  - M & M Medical Center, Inc, Miami, Florida
  - Med Research Of Florida, LLC, Miami, Florida
  - Research Physicians Network Alliance, Miami Beach, Florida
  - G & I Medical Research LLC, Miami Lakes, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Southwest Florida Research, LLC, Naples, Florida
  - BayCare Medical Group, New Port Richey, Florida
  - The Heart & Vascular Institute of Florida, New Port Richey, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - Harmony Clinical Research, Inc., North Miami Beach, Florida
  - Florida Hospital, Orlando, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Aba Family Medicine, LLC, Ormond Beach, Florida
  - Millennium Research, Ormond Beach, Florida
  - Ribo Research, LLC dba Peninsula Research, Ormond Beach, Florida
  - A and R Research Group LLC, Pembroke Pines, Florida
  - Research Physicians Network Alliance, Pembroke Pines, Florida
  - South Broward Research, Pembroke Pines, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - DBC Research, Pembroke Pines, Florida
  - Cardiology Consultants, Pensacola, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Clinical Research of Central Florida, Plant City, Florida
  - Clinical Research of Florida, Plant City, Florida
  - Jeffrey D Greff,MD, Plantation, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Cardiovascular Center Of Sarasota, Sarasota, Florida
  - Heart & Vascular Center Research, Sarasota, Florida
  - Intercoastal Medical Group (Drug Shipment Address and Administrative), Sarasota, Florida
  - The Office of Bridget Bellingar, DO, Seminole, Florida
  - Meridien Research, St. Petersburg, Florida
  - Advance Medical Research, St. Petersburg, Florida
  - Vita Health & Medical Center, Inc./Concept Clinical Trials, LLC, Tamarac, Florida
  - Interventional Cardiac Consultants, Trinity, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Cleveland Clinic Cardiology Associates, West Palm Beach, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta Center For Medical Research, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Rockdale Medical Research Associates, Conyers, Georgia
  - Georgia Heart Specialists, LLC, Covington, Georgia
  - Neurostudies.net, LLC, Decatur, Georgia
  - Alta Pharmaceutical Research Center, Dunwoody, Georgia
  - In-Quest Medical Research, LLC, Norcross, Georgia
  - Atlanta Center for Clinical Research / Internal Medicine, Roswell, Georgia
  - Dr. B. Abraham, P.C., Snellville, Georgia
  - Georgia Clinical Research, LLC, Snellville, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Elite Clinial Trials, LLLP, Blackfoot, Idaho
  - Elite Clinical Trials (Additional Administrative Room / Exam Rooms), Blackfoot, Idaho
  - St. Luke's Idaho Cardiology Associates, Caldwell, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Saltzer Medical Group, PA, Nampa, Idaho
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Clinical Research Advantage, Inc./Michigan Avenue Internists, Chicago, Illinois
  - Apex Medical Research, AMR, Inc., Chicago, Illinois
  - Clinical Research Advantage,Inc./Medical and Procedural Specilaists of Illinois, Chicago, Illinois
  - Evanston Premier Healthcare Research, LLC, Evanston, Illinois
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - Heart Care Centers of Illinois, Mokena, Illinois
  - Advanced CardioVascular Consultants, Rock Island, Illinois
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - Investigative Clinical Research of Indiana, LLC, Elwood, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Clinical Research Advantage, Inc., Evansville, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Clinical Research Advantage, Inc. / Family Medicine Associates, Evansville, Indiana
  - Deaconess Clinic Mt. Pleasant, Evansville, Indiana
  - American Health Network of Indiana LLC, Franklin, Indiana
  - American Health Network of Indiana LLC, Greenfield, Indiana
  - American Health Network of Indiana, LLC, Muncie, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Clinical Research Advantage, Inc., Council Bluffs, Iowa
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Iowa-College of Public Health-Preventive Intervention Center, Iowa City, Iowa
  - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - Hutchinson Clinic, P.A, Hutchinson, Kansas
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Midwest Heart & Vascular Specialists, LLC, Overland Park, Kansas
  - Women's & Family Care D.B.A. GTC Research, Shawnee Mission, Kansas
  - Women's & Family Care, LLC D.B.A GTC Research, Shawnee Mission, Kansas
  - Women's & Family Care, LLC D.B.A. GTC Research, Shawnee Mission, Kansas
  - Central Cardiology Associates Research, Elizabethtown, Kentucky
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - L-MARC, Louisville, Kentucky
  - Research Integrity, LLC., Owensboro, Kentucky
  - Grace Research, LLC, Bossier City, Louisiana
  - Avant Research Associates, LLC, Crowley, Louisiana
  - Centex Studies, Lake Charles, Louisiana
  - Imperial Health, LLP, Lake Charles, Louisiana
  - American Clinical Research, LLC, Marrero, Louisiana
  - West Jefferson Heart Clinic of Louisiana New Orleans Physician Services, Inc., Marrero, Louisiana
  - Clinical Trials of America LA, Monroe, Louisiana
  - KAMP Medical Research Inc., Natchitoches, Louisiana
  - Clinical and Translation Research Center (CTRC) University Medical Center of New Orleans, Diagnostic, New Orleans, Louisiana
  - Section of Nephrology and Hypertension, LSU Health Sciences Center-New Orleans, New Orleans, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Acadia Clinical Research, LLC, Bangor, Maine
  - Acadia Clinical Research, Bangor, Maine
  - Cranbrook Cardiology Research Associates, Cape Elizabeth, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - MedStar Cardiology Associates, Annapolis, Maryland
  - MedStar Chesapeake CardioVascular Associates, Baltimore, Maryland
  - MedStar Union Memorial Heart Specialists, Baltimore, Maryland
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Overlea Personal Physicians, Baltimore, Maryland
  - Shahid Saeed, MD, PC, Baltimore, Maryland
  - Maryland Heart Associates, LLC, Glen Burnie, Maryland
  - Lutherville Personal Physicians, Lutherville, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - MetroWest Medical Center - Pharmacy Department, Framingham, Massachusetts
  - MetroWest Medical Center Research Clinic, Framingham, Massachusetts
  - MetroWest Medical Center, Framingham, Massachusetts
  - ActivMed Practices and Research, Inc., Methuen, Massachusetts
  - Charles River Medical Associates, Natick, Massachusetts
  - Endeavor Medical Research, Alpena, Michigan
  - St. Joseph Mercy Health System (Drug shipment Only), Ann Arbor, Michigan
  - University of Michigan - Domino Farms, Ann Arbor, Michigan
  - Quest Research Institute, Bingham Farms, Michigan
  - IHA Chelsea Family & Internal Medicine, Chelsea, Michigan
  - Healthy Heart Cardiology, Grandville, Michigan
  - Westside Family Medical Center, Pc, Kalamazoo, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Sparrow Thoracic & Cardiovascular Institute, Lansing, Michigan
  - Detroit Clinical Research Center, PC, Livonia, Michigan
  - MidMichigan Medical Center Midland, Midland, Michigan
  - Michigan Cardio Vascular Institute, Saginaw, Michigan
  - Tri-County Research, Inc., Sterling Heights, Michigan
  - Medical Research Associates, Inc., Traverse City, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Arcturus Healthcare, PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Michigan Heart & Vascular Institute, Ypsilanti, Michigan
  - Duluth Clinic, dba Essentia Health Duluth Clinic Investigational Drug Room, Duluth, Minnesota
  - St. Mary's Medical Center dba Essentia Health St. Mary's Medical Center, Duluth, Minnesota
  - St. Mary's Medical Center, Duluth, Minnesota
  - The Duluth Clinic, Ltd., Duluth, Minnesota
  - Radiant Research, Inc., Edina, Minnesota
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Allina Health System, dba Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Lillehei Clinical Research Unit, University of Minnesota, Minneapolis, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - HealthEast St. Joseph's Hospital inpatient Pharmacy, Saint Paul, Minnesota
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Missouri Cardiovascular Specialists, LLP, Columbia, Missouri
  - Saint Luke's Lipid and Diabetes Research Center, Kansas City, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Mercy Research, St Louis, Missouri
  - Glacier View Research Institute, Cardiology, Kalispell, Montana
  - Montana Medical Research Inc., Missoula, Montana
  - Bryan Heart, Lincoln, Nebraska
  - Creighton Diabetes Research Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - AB Clinical Trials, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Clinical Research Advantage, Inc., Las Vegas, Nevada
  - John V. Bernard, MD dba Wellness and Research Center, Belvidere, New Jersey
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Lourdes Cardiology Services, Cherry Hill, New Jersey
  - USMA Clinical Research, Elizabeth, New Jersey
  - Lourdes Cardiology Services, Hammonton, New Jersey
  - NJ Heart, Linden, New Jersey
  - Arysmed LLC, Lodi, New Jersey
  - Amici Clinical Research, LLC, Martinsville, New Jersey
  - Rutgers Biomedical and Health Sciences-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cardiac & Endovascular Associates, Ridgewood, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - TLB Research LLC, Trenton, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Westwood Cardiology Associates, P.A., Westwood, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Sorin Medical, P.C., Brooklyn, New York
  - NY Total Medical Care, PC, Brooklyn, New York
  - NY Scientific, Brooklyn, New York
  - Buffalo Heart Group, Llp, Buffalo, New York
  - NYU Hudson Valley Cardiology, Cortlandt Manor, New York
  - Scott Research,Inc, Laurelton, New York
  - SJH Cardiology Associates, Liverpool, New York
  - Long Island Heart Associates, Mineola, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Manhattan Medical Research Practice, New York, New York
  - Peters Medical Research NY, LLC, New York, New York
  - Weill Cornell Medical College, New York, New York
  - DiGiovanna Institute for Medical Education And Research, North Massapequa, New York
  - Hudson Valley Cardiovascular Practice, PC, Poughkeepsie, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Institute for Clinical Studies, Rosedale, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Central New York Cardiology, Utica, New York
  - Great Lakes Medical Research, Westfield, New York
  - Buffalo Medical Group, Williamsville, New York
  - Novant Health Clinical Research, Charlotte, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Sensenbrenner Primary Care, Charlotte, North Carolina
  - NC Heart and Vascular, Clayton, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - Carolina Cardiology Cornerstone, High Point, North Carolina
  - Clinical Trials of America- NC, LLC, Lenoir, North Carolina
  - Research Institute of the Carolinas of Piedmont Healthcare, PA, Mooresville, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Eastern Nephrology Associates, New Bern, North Carolina
  - Boice Willis Clinic, Rocky Mount, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - NC Heart and Vascular Research, Smithfield, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Wake Forest University Health Sciences Institutional Review Board, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Radiant Research, Inc, Akron, Ohio
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Dayton Heart Center, Dayton, Ohio
  - Premier Health Specialists, Inc. (dba Dayton Heart Center), Dayton, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Delaware Research Group, LLC, Delaware, Ohio
  - North Ohio Heart Center (Administrative Only), Elyria, Ohio
  - North Ohio Heart Center, Elyria, Ohio
  - North Ohio Heart Center, Lorain, Ohio
  - SV Research LLC, Marion, Ohio
  - Office of Daniel G. Williams, MD, Perrysburg, Ohio
  - North Ohio Heart Center, Inc., Sandusky, Ohio
  - ProMedica Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Mercy Health Youngstown, LLC d/b/a St. Elizabeth Youngstown Hospital, Youngstown, Ohio
  - LION Research, Norman, Oklahoma
  - COR Clinical Research LLC, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Physicians, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Integrated Medical Research PC, Ashland, Oregon
  - Hillsboro Cardiology, PC, Hillsboro, Oregon
  - Portland Preventive Cardiology LLC, Portland, Oregon
  - Abington Hosptial, Abington, Pennsylvania
  - Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Doylestown Cardiology Associates - VIAA, Doylestown, Pennsylvania
  - Doylestown Health Cardiology, a division of Doylestown Health Physicians, Doylestown, Pennsylvania
  - Amh/Feasterville Family Health Care Center, Feasterville-Trevose, Pennsylvania
  - Greater Pittsburgh Vascular, Jefferson Hills, Pennsylvania
  - Detweiler Family Medicine and Associates, PC, Lansdale, Pennsylvania
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Family Medical Associates, Levittown, Pennsylvania
  - Mercer Bucks Cardiology, Newtown, Pennsylvania
  - Philadelphia Health Associates-Adult Medicine, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - SFM Clinical Trials, Inc., Scotland, Pennsylvania
  - Fay-West Family Practice, Scottdale, Pennsylvania
  - Grand View - Lehigh Valley Health Services, Buxmont Cardiology Division, Sellersville, Pennsylvania
  - Montgomery Medical, Inc., Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Berks Cardiologists, Ltd., Wyomissing, Pennsylvania
  - Coastal Cardiology, Charleston, South Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - The Diabetes Center, LLC, Murrells Inlet, South Carolina
  - Black Hills Cardiovascular-Regional Health Research, Rapid City, South Dakota
  - Mid-Cumberland Infectious Disease Consultants, PLC, Clarksville, Tennessee
  - Collierville Medical Specialists, Collierville, Tennessee
  - Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - PMG Research,Inc d/b/a PMG Research of Knoxville, Knoxville, Tennessee
  - Cardiovascular Research of Knoxville, Knoxville, Tennessee
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Baptist Memorial Medical Group, Inc., Memphis, Tennessee
  - The Green Clinic, PC, Memphis, Tennessee
  - Southwind Medical Specialists, Memphis, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Trinity Clinical Research, LLC, Tullahoma, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - Arlington Family Research Center, Inc., Arlington, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Austin Heart, PLLC, Austin, Texas
  - Aztec Medical Research, LLC, Channelview, Texas
  - Corsicana Medical Research, PLLC, Corsicana, Texas
  - Protenium Clinical Research, LLC, Dallas, Texas
  - VA North Texas Health Care System - Dallas VAMC, Dallas, Texas
  - Baylor Heart and Vascular Institute, Dallas, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Radiant Research, Inc., Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Doctors Hospital At Renaissance, Edinburg, Texas
  - Amir Malik Research, Fort Worth, Texas
  - The Medical Group Of Texas, Fort Worth, Texas
  - Rockwood Medical Clinic, Fort Worth, Texas
  - San Gabriel Clinical Research, LLC, Georgetown, Texas
  - East Texas Cardiology PA, Houston, Texas
  - Spring Clinical Research, Houston, Texas
  - Med Tech Research, LP, Houston, Texas
  - Prime Care Medical Group, Houston, Texas
  - Associates in Medicine, PA, Houston, Texas
  - Alan S. Hoffman, M.D., Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Investigational Product Shipment Address TO: Investigational Drug Services (IDS),, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Northwest Houston Cardiology, Houston, Texas
  - Texas Center For Drug Development, Inc., Houston, Texas
  - Private Practice Leadership, LLC, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - South Texas Cardiovascular Consultants, PLLC, Kerrville, Texas
  - Caprock Cardiac Center Research Institute Inc., Lubbock, Texas
  - Midland Clinical Research Center, Midland, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - North Hills Medical Research, Inc., North Richland Hills, Texas
  - Grace Research, LLC, Palestine, Texas
  - Med-Olam Clinical Research, Pasadena, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Austin Institute for Clinical Research,Inc., Pflugerville, Texas
  - Centex Studies, Inc, Pharr, Texas
  - Legacy Heart Center, Plano, Texas
  - South Texas Cardiovascular Consultants, PLLC, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Southwest Clinic, San Antonio, Texas
  - Victorium Clinical Research, San Antonio, Texas
  - Bandera Family Health Care, LLC, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, LLC (NECRSA, LLC), Schertz, Texas
  - Acacia Medical Research Institute, LLC, Sugar Land, Texas
  - IP + Dry ice deliveries Sugar Lakes Family Practice, Sugar Land, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Admin & Storage only:Northwest Heart Center, Tomball, Texas
  - Northwest Heart Center, Tomball, Texas
  - Northwest Houston Clinical Research, PLLC, Tomball, Texas
  - Victoria Heart and Vascular Center, PA, Victoria, Texas
  - Utah Cardiology, PC, Bountiful, Utah
  - Utah Cardiology, P.C., Layton, Utah
  - Paramount Medical Care, Ogden, Utah
  - Aspen Clinical Research LLC, Orem, Utah
  - Revere Health, Provo, Utah
  - Optimum Clinical Research, Inc., Salt Lake City, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Holladay Family Practice, Salt Lake City, Utah
  - Heart Center at St. Mark's Hospital, Salt Lake City, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Clinical Research Institute of Northern Virginia, Burke, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Seven Corners Medical Research Center, Falls Church, Virginia
  - Heart Care Associates, P.C., Hopewell, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - Chippenham and Johnston Willis Hospitals, Inc. dba CJW Medical Center, Richmond, Virginia
  - Retreat Cardiology LLC, dba Cardiology Associates of Richmond, Richmond, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
  - Hampton Roads Center for Clinical Research, Suffolk, Virginia
  - Office of Daniel W. Gottlieb, MD, PS, Burien, Washington
  - Premier Clinical Research, Spokane, Washington
  - Universal Research Group, LLC, Tacoma, Washington
  - Walla Walla Clinic, Walla Walla, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - Exemplar Research Inc, Fairmont, West Virginia
  - Prevea Clinic, Inc., Green Bay, Wisconsin
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
  - Waukesha Heart Foundation, Waukesha, Wisconsin
- Argentina (43):
  - Instituto de Investigaciones Clinicas Bahia Blanca, Bahía Blanca, Buenos Aires
  - Hospital Italiano Regional del Sur, Bahía Blanca, Buenos Aires
  - CIPREC - Centro de Investigacion y Prevencion Cardiovascular S.A., C.a.b.a., Buenos Aires
  - Hospital Britanico De Buenos Aires, Ciudad Autonoma de B. Aires, Buenos Aires
  - Investigaciones Medicas IMOBA S.R.L., Ciudad Autonoma de Buenos Aires, Buenos Aires
  - CEDIC - Consultorios Medicos, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Clinica Coronel Suarez S.A., Coronel Suárez, Buenos Aires
  - Framingham Centro Medico, La Plata, Buenos Aires
  - CIMeL CHAHIN CHAHIN S.A., Lanús Este, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - DIM Clinica Privada, Ramos Mejía, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - STAT Research S.A., C.a.b.a, Buenos Aires F.D.
  - Consultorios Asociados de Endocrinologia e Investigacion Clinica Aplicada, C.a.b.a, C.a.b.a.
  - Clinica Privada de Especialidades Medicas, Villa María, Córdoba Province
  - CIPADI Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz, Mendoza Province
  - IMEP Instituto Medico Elsa Perez, Ciudadela, PCIA de Buenos Aires
  - Instituto Medico Aguero, Morón, PCIA de Buenos Aires
  - Cordis - Instituto del Corazon, Resistencia, PCIA de Chaco
  - Hospital de Alta Complejidad "Pte. Juan Domingo Peron", Formosa, PCIA de Formosa
  - Hospital Provincial Dr. Jose Maria Cullen, Santa Fe, PCIA de Santa FE
  - Centro De Investigaciones Clinicas Del Litoral S.R.L., Santa Fe, PCIA de Santa FE
  - Cedir S.A - Centro De Diagnostico Y Rehabilitacion S.A., Santa Fe, PCIA de Santa FE
  - Centro Modelo de Cardiologia, San Miguel de Tucumán, PCIA de Tucuman
  - Instituto de Hematologia y Medicina Clinica "Dr. Ruben A. Davoli", Rosario, Pcia. de Santa FE
  - Instituto Medico Ceniclar - Central De Investigaciones Clinicas Argentina - Sanatorio De La Mujer, Rosario, Santa Fe Province
  - Centro Medico CCBR Tucuman, San Miguel de Tucumán, Tucumán Province
  - Universidad Maimonides, Buenos Aires
  - Centro de Investigacion: AXISMED S.R.L., Buenos Aires
  - Cicemo - Consultorio de Investigaciones Clinicas E.M.O. S.R.L., Ciudad Autonoma de B. Aires
  - Instituto Cardiovascular De Buenos Aires, Ciudad Autonoma de B. Aires
  - Instituto de Cardiologia de Corrientes "Juana Fca. Cabral", Corrientes
  - ILAIM Instituto Latinoamericano de Investigaciones Medicas, Córdoba
  - Clinico Chutro SRL, Córdoba
  - Centro de Investigaciones Clinicas "Instituto del Corazon", Córdoba
  - Clinica Privada Colombo, Córdoba
  - Instituto Medico DAMIC S.R.L., Córdoba
  - Centro Medico Luquez, Córdoba
  - IPAC Caraffa, Córdoba
  - Hospital Central de Mendoza, Mendoza
  - Cordis S.A., Salta
  - Centro Cardiovascular Salta, Salta
  - Instituto Cardiovascular San Luis A.E., San Luis
- Australia (25):
  - Boden Institute of Obesity, Nutrition, Exercise and Eating Disorders, Camperdown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Central Coast Neurosciences Research, Erina, New South Wales
  - Central Coast Local Health District, Gosford Hospital, Gosford, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Holy Spirit Northside Private Hospital Limited, Chermside, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Core Research Group Pty Ltd, Milton, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Austrials Pty Ltd, Sherwood, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Adelaide Medical Research, Ashford, South Australia
  - SA Heart, Ashford, South Australia
  - Southern Adelaide Diabetes and Endocrine Service, Daws Park, South Australia
  - Department of Cardiology, Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Heart and Vascular Research, Fullarton, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Eastern Health - Box Hill Hospital, Box Hill, Victoria
  - The Northern Hospital, Epping, Victoria
  - Barwon Health-The Geelong Hospital, Geelong, Victoria
  - Austin Health - Heidelberg Repatriation Hospital, Heidelberg West, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - HPS Pharmacies, Joondalup, Western Australia
  - Joondalup Cardiovascular Trials Foundation Inc., Joondalup, Western Australia
- Belgium (34):
  - VZW Algemeen Ziekenhuis KLINA, Brasschaat, Antwerpen
  - AZ Sint-Maarten, Mechelen, Antwerp
  - Algemeen Stedelijk Ziekenhuis, Aalst, Oost-vlaanderen
  - Az Sint Blasius, Dendermonde, Oost-vlaanderen
  - AZ Sint Lucas Gent, Ghent, Oost-vlaanderen
  - Universitair Ziekenhuis Gent, Ghent, Oost-vlaanderen
  - Az Glorieux, Ronse, Oost-vlaanderen
  - AZ Nikolaas, Campus Moerland, Sint-Niklaas, Oost-vlaanderen
  - AZ Groeninge-Campus Loofstraat, Kortrijk, West-vlaanderen
  - Az Damiaan, Ostend, West-vlaanderen
  - ZNA Campus Middelheim, Antwerp
  - Imeldaziekenhuis Bonheiden, Bonheiden
  - A.Z. St.Jan AV Brugge, Bruges
  - University Hospital Brussels - Centrum voor hart- en vaatziekten, Brussels
  - University Hospital Brussels- Diabeteskliniek, Brussels
  - Private Practice 'Cardiovascular Detection Center', De Pinte
  - ZOL Campus Sint-Jan, Genk
  - AZ Maria Middelares, Ghent
  - Grand Hopital de Charleroi, Site St-Joseph, Gilly
  - Hygeia, Hasselt
  - Jessa Ziekenhuis, Hasselt
  - Sint-Franciskusziekenhuis, Heusden-Zolder
  - Centre Hospitalier Regional de Huy, Huy
  - Jan Yperman Ziekenhuis, Cardiology, Ieper
  - Centre Hospitalier De Jolimont - Lobbes, La Louviere (Haine-Saint-Paul)
  - Centre Hospitalier de Jolimont-Lobbes, La Louviere (Haine-Saint-Paul)
  - University hospitals Leuven - Neurology department, Leuven
  - University hospitals Leuven, Leuven
  - Centre Hospitalier Universitaire (CHU) de Liege, Liège
  - Huisartsenpraktijk Medilink, Linkebeek
  - Huisartsenpraktijk Luc Capiau, Massemen
  - C.H.U. Ambroise Pare, Mons
  - Mariaziekenhuis vzw, Overpelt
  - Dr. Luc De Wolf - Private Practice, Tienen
- Brazil (29):
  - Centro de Pesquisas em Diabetes e Doencas Endocrino-Metabolicas Ltda, Fortaleza, Ceará
  - Fundacao Bahiana De Cardiologia, Salvador, Estado de Bahia
  - HBA S/A ASSISTENCIA MEDICA E HOSPITALAR-Hospital da Bahia, Salvador, Estado de Bahia
  - Covance Central Laboratory Services, Indianapolis, Indiana
  - CARDSEARCH/CARDRESEARCH - Cardiologia Assistencial e de Pesquisa LTDA, Belo Horizonte, Minas Gerais
  - Sociedade Hospitalar Angelina Caron/Hospital e Maternidade Angelina Caron, Campina Grande do Sul, Paraná
  - Hospital Santa Casa de Curitiba, Curitiba, Paraná
  - Quanta Diagnostico e Terapia / Medicina Nuclear Alto da XV, Curitiba, Paraná
  - Nucleo de Pesquisa Clínica, Curitiba, Paraná
  - Universidade Federal do Para - Hospital Universitario Joao de Barros Barreto, Belém, Pará
  - Centro de Pesquisas Medicas Basica e Clinica LTDA, Recife, Pernambuco
  - Hospital Agamenon Magalhaes, Recife, Pernambuco
  - CCBR Brasil - Centro de Pesquisa e Analises Clinicas LTDA, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitario - Associacao Educadora Sao Carlos - AESC, Canoas, Rio Grande do Sul
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus/Associacao Educadora Sao Carlos AESC / IMV - Instituto de Medicina Vascular, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia do Rio Grande do Sul / Fundacao Universitaria de Cardiologia, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus - Instituto do Cancer, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus-Associacao Educadora de Sao Carlos-AESC/IMV - Instituto de Medicina Vascular, Porto Alegre, Rio Grande do Sul
  - Mae de Deus - Centro de Oncologia Radioterapica (COR), Porto Alegre, Rio Grande do Sul
  - Hospital Santa Isabel, Blumenau, Santa Catarina
  - Loema Medicina e Bem Estar- Centro Especializado em Cardiologia Ltda., Campinas, São Paulo
  - CAEP - Centro Avançado de Estudos e Pesquisas Ltda., Campinas, São Paulo
  - IMC - Instituto de Molestias Cardiovasculares/Equipamentos Cardiovasculares Rio Preto Ltda, São José do Rio Preto, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo (HC-FMUSP), São Paulo, São Paulo
  - CARDSEARCH/CARDRESEARCH - Cardiologia Assistencial e de Pesquisa LTDA, Minas Gerais
  - CPClin- Centro de Pesquisas Clinicas Ltda./Clinica Dr. Freddy Goldberg Eliaschewitz, São Paulo
  - FGM-Clinica Paulista de Doencas Cardiovasculares, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica e Servicos Medicos Ltda, São Paulo
- Canada (66):
  - LMC Diabetes & Endocrinology (Calgary), Calgary, Alberta
  - Foothills Hospital/University of Calgary, Calgary, Alberta
  - Nanji Professional Corporation, Calgary, Alberta
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - Kelowna Cardiology Associates, Kelowna, British Columbia
  - Dr. Raymond Dong Inc., Surrey, British Columbia
  - Dr. Richard Bon Inc. & Dr. Adam Yeung Inc., Surrey, British Columbia
  - Dr. Stephen S. Cheung Inc., Surrey, British Columbia
  - SMH Cardiology Clinical Trials, Surrey, British Columbia
  - Dr. Dante E. Manyari Inc., Surrey, British Columbia
  - Dr. Stephanie Au, Inc., Surrey, British Columbia
  - Dr. Stephen Pearce Inc. & Dr. Peter K.H. Tan Inc., Surrey, British Columbia
  - SMH Cardiology Clinical Trials Inc, Surrey, British Columbia
  - Dr. Adam Yeung Inc., Surrey, British Columbia
  - Dr. Michael Kanakos Inc., Surrey, British Columbia
  - Dr. Kapil M. Bhagirath Medical Services Corporation, Surrey, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Discovery Clinical Services Ltd., Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Cardiology Research Associates of New Brunswick, Saint John, New Brunswick
  - Health Sciences Centre, St. John's, NF
  - Health Science Centre, St. John's, NF
  - LMC Diabetes & Endocrinology (Brampton), Brampton, Ontario
  - Aviva Clinical Trial Group Inc., Burlington, Ontario
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - Philippe R. Beaudry Medicine Professional Corporation, Burlington, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Vizel Cardiac Research - Saul Vizel Professional Medicine Corporation, Cambridge, Ontario
  - Moran Medical Centre, Collingwood, Ontario
  - C & L Research, Fort Erie, Ontario
  - Brian Y.L. Wong Medicine Professional Corporation, Greater Sudbury, Ontario
  - Parkdale Medical Centre, Hamilton, Ontario
  - Stroke Prevention & Atherosclerosis Research Centre (SPARC), London, Ontario
  - Western University - WCPHFM, London, Ontario
  - LMC Diabetes & Endocrinology (Markham), Markham, Ontario
  - Newmarket Cardiology Research Group, Newmarket, Ontario
  - LMC Clinical Research Inc. (Oakville), Oakville, Ontario
  - The Office of Dr. James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - Scarborough Cardiology Research Associates Inc., Scarborough Village, Ontario
  - Canadian Centre for Research on Diabetes, Smiths Falls, Ontario
  - LMC Diabetes & Endocrinology (Thornhill), Thornhill, Ontario
  - JJ Dig Research LTD, Toronto, Ontario
  - Canadian Phase Onward, Inc., Toronto, Ontario
  - LMC Diabetes & Endocrinology (Bayview), Toronto, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Dr. Mohan Babapulle Medicine Professional Cooperation, Waterloo, Ontario
  - Dr. Louis Yao, MD Office of, Weston, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Q & T Research Chicoutimi, Chicoutimi, Quebec
  - Q&T Recherche Outaouais Inc., Gatineau, Quebec
  - Omnispec Recherche Clinique Inc., Mirabel, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Diex Research Montreal, Inc., Montreal, Quebec
  - Recherche Clinique Sigma inc, Québec, Quebec
  - Clinique des maladies lipidiques de Quebec, Québec, Quebec
  - Centre integre de sante et de services sociaux de Lanaudiere (CISSSL), Saint-Charles-Borromée, Quebec
  - CISSS des Laurentides-Point de Service de St-Jerome- Comite d'ethique de la recherche, Saint-Jérôme, Quebec
  - St-Jerome Medical Research Inc., Saint-Jérôme, Quebec
  - LMC Clinical Research Inc. (Montreal), Saint-Laurent, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke - Hotel-Dieu, Sherbrooke, Quebec
  - Centre Integre de Sante et de services sociaux de Chaudiere-Appalaches (CISSA-CA) -, St-Georges, Beauce, Quebec
  - C.I.C. Mauricie Inc., Trois-Rivières, Quebec
- Chile (9):
  - Corporacion de Beneficencia Osorno, Osorno, Los Lagos Region
  - Centro de Investigacion Clínica del Sur, Temuco, Región de la Araucanía
  - Biomedica Research Group, Providencia Santiago, Santiago Metropolitan
  - CICAB, Santiago, Santiago Metropolitan
  - Servicios Medicos Godoy, Santiago, Santiago Metropolitan
  - SMOLAM, Santiago, Santiago Metropolitan
  - Complejo Asitencial Dr. Sotero del Rio, Santiago, Santiago Metropolitan
  - Quantum Research, Puerto Varas
  - Hospital y CRS El Pino, Santiago
- Colombia (20):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Rodrigo Botero S.A.S, Medellín, Antioquia
  - Centro de Investigacion Clinica Avanzada y Multidisciplinaria CICLAM, Medellín, Antioquia
  - Centro de Medicina del Ejercicio y Rehabilitacion Cardiaca S.A. CEMDE S.A., Medellín, Antioquia
  - Clinica de la Costa LTDA, Barranquila, Atlántico
  - Centro Cientifico Asistencial Jose Luis Accini S.A.S., Barranquilla, Atlántico
  - Corazon Ips S.A.S., Barranquilla, Atlántico
  - Corozan Ips Sas, Barranquilla, Atlántico
  - Fundacion del Caribe para la Investigacion Biomedica - Fundacion BIOS, Barranquilla, Atlántico
  - Asociacion IPS Medicos Internistas de Caldas, Manizales, Caldas Department
  - MedPlus Medicina Prepagada S.A., Bogota D.C., Cundinamarca
  - Solano & Terront Servicios Medicos Ltda-Establecimiento Comercial UNIENDO, Bogota D.C., Cundinamarca
  - Dexadiab Servicios Medicos LTDA, Bogota D.C, Cundinamarca
  - Caja de Compensacion Familiar CAFAM, Sede Centro de Atencion en Salud CAFAM FLORESTA, Bogota D.C, Cundinamarca
  - Hospital Universitario San Ignacio, Bogota D.C, Cundinamarca
  - Instituto de Investigacion Endocrinologia y Prevencion Metabolica - ENDOCARE LTDA., Bogota D.C, Cundinamarca
  - Centro de Diagnostico Cardiologico LTDA., Cartagena, Departamento de Bolívar
  - Instituto del Corazon de Bucaramanga S.A., Bucaramanga, Santander Department
  - Fundación Cardiovacular de Colombia - Instituto del Corazón de Floridablanca, Floridablanca, Santander Department
  - Fundacion Reina Isabel, Cali, Valle del Cauca Department
- Czechia (30):
  - FREMLOVA APHOTECA s.r.o., Litovel, Czech Republic
  - BENU Lekarna, Pardubice, Czech Republic
  - EDUMED s.r.o., Broumov, Královéhradecký kraj
  - Edumed S.R.O., Jaroměř, Královéhradecký kraj
  - Kardiologicka ambulance, Trutnov, Královéhradecký kraj
  - Lekarna na Poliklinice, Trutnov, Královéhradecký kraj
  - MUDr. Jan Vrkoc s.r.o., Ostrava, Moravskoslezský kraj
  - Pv-Kardiologie S.R.O., Pardubice, Pardubický kraj
  - Kardiologicka Ambulance, Brno, South Moravian
  - CCBR Czech Brno, s.r.o., Brno
  - DIKa centrum s.r.o., Kardiologicka a interni ambulance, Havířov
  - Fakultni nemocnice Hradec Kralove, III. Interni gerontometabolicka klinika, Hradec Králové
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Kardio interna s.r.o., Litovel
  - Fakultni Nemocnice Olomouc, Olomouc
  - CCBR Czech a.s., Pardubice
  - Kardiologie Plzen s.r.o., Pilsen
  - Fakultni poliklinika Vseobecne fakultni nemocnice v Praze, Prague
  - CCBR Czech Prague, s.r.o, Prague
  - Centrum kardiovaskularni prevence 1. LF UK a TN, Prague
  - Kardiologie a interni lekarstvi, Prague
  - NEFROMED, s.r.o., Prague
  - Interna a kardiologie s.r.o., Rožnov pod Radhoštěm
  - Nemocnice Pardubickeho kraje, a.s., Svitavska nemocnice, Svitavy
  - Vseobecna kardiologicka ambulance s.r.o., Tábor
  - Lekarna U Nemocnice, Tábor
  - Lekarna Hradebni s.r.o., Uherské Hradiště
  - MUDr. Antonin Dufka, kardiologicka ambulance, Uherské Hradiště
  - MUDr. Nina Zemkova s.r.o., Uherské Hradiště
  - KIGE s.r.o., Znojmo
- Denmark (26):
  - Sygehus Sonderjylland Aabenraa, Aabenraa
  - Aalborg Universitetshospital, Lipidklinikken, Aalborg
  - CCBR Aalborg, Aalborg
  - Aarhus Universitetshospital Skejby, Hjertesygdomme ¿ Klinisk Forskning, Aarhus
  - Aarhus Universitetshospital, Aarhus N
  - CCBR Ballerup, Ballerup Municipality
  - Bispebjerg og Frederiksberg Hospital, Copenhagen NV
  - Rigshospitalet, Copenhagen Oe
  - Sydvestjysk Sygehus, Esbjerg
  - Frederiksberg Hospital, Frederiksberg
  - Glostrup Hospital, Glostrup Municipality
  - Herlev Universitetshospital, Kardiologisk afdeling S, Herlev
  - Regionshospitalet Herning, Herning
  - Hillerod Hospital, Hillerød
  - Hvidovre Universitetshospital, Hjerte-lungemedicinsk afdeling, Hvidovre
  - Kolding Sygehus, Kolding
  - Amager Hospital, København S
  - Region Sjaelland Sygehus Nord, Koge Sygehus, Køge
  - Nykobing F. Sygehus-Medicinsk afdeling, Nykøbing Falster
  - Region Sjaelland Naestved Sygehus, Næstved
  - Regionshospitalet Randers, Randers
  - Regionshospitalet Silkeborg, Hjerte Projektkontor, Silkeborg
  - Slagelse Sygehus, Slagelse
  - Svendborg Sygehus, Svendborg
  - CCBR Vejle, Vejle
  - Hospitalsenheden Midt, Regionshospital Viborg, Viborg
- Finland (21):
  - Linnan Klinikka Oy, Hämeenlinna
  - Mehilainen Toolo, Helsinki
  - Helsinki University Central Hospital, Helsinki
  - Helsingin yliopistollinen keskussairaala, Sisaetaudit ja kuntoutus, Biomedicum 2U, Helsinki
  - Ita-Suomen laakarikeskus Oy, Joensuu
  - Studycor Oy, Jyväskylä
  - Laeaekaerikeskus Aava Kerava, Kerava
  - Menoa oy, Kinkomaa
  - Kokkolan Keskussairaala, Kokkola
  - Mewell liikuntaklinikka, Kotka
  - Itae-Suomen Laeaekaeritalo Oy, Kuopio
  - Terveystalo Kuopio, Kuopio
  - Oulu Mentalcare Oy, Oulu
  - Terveystalo Oulu, Diapolis, Oulu
  - Oulu University Hospital, Oulu
  - Porin Laakaritalo Oy, Pori
  - Terveystalo Siilinjarvi, Siilinjärvi
  - FinnMedi Oy, Tampere
  - Terveystalo Pulssi, Turku
  - Turku University Hospital, Turku
  - Vantaan Tutkimuskeskus, Vantaa
- France (23):
  - CHU Jean Minjoz Cardiologie, Besançon
  - Centre Hospitalier De Bourg En Bresse - Hopital Fleyriat, Bourg-en-Bresse
  - CHU de Caen, Caen
  - Centre Hospitalier de Cannes- Service de Cardiologie, Cannes
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Scp Cardiovasculaire De L'Est, Essey-lès-Nancy
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Hopital La Louviere, Lille
  - Centre Hospitalier Saint Philibert, Lomme
  - Hopital Cardiovasculaire Et Pneumologique Louis Pradel, Lyon
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHU de Nantes - Hopital Nord Laennec, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - CHU Caremeau, Nîmes
  - Centre Hospitalier de PAU, Pau
  - Hopital Cardiologique, Pessac
  - CHU de Poitiers, Poitiers
  - CHU de Renes Hopital de Pontchaillou, Rennes
  - CHU de Toulouse, Toulouse
  - Hopital Guy Chatiliez, Tourcoing
  - Hopital Trousseau, Tours
  - Centre Hospitalier (CH) de Valenciennes, Valenciennes
  - Polyclinique Vauban, Valenciennes
- Germany (70):
  - Universitaets Herzzentrum Freiburg Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Medizinische Universtatsklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Ze:ro Arztpraxen, Mannheim, Baden-Wurttemberg
  - Gemeinschaftspraxis im Altstadt Carree, Fulda, Hesse
  - Klinische Forschung Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Zentrum Klinische Studien Neuwied (ZKSN), Neuwied, Rhineland-Palatinate
  - Gemeinschaftspraxis Schwabenheim, Schwabenheim, Rhineland-Palatinate
  - Klinikum Altenburger Land Gmbh, Altenburg
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Forschungszentrum Dr. med Irma Schoell, Bad Homburg
  - Institut fuer Klinische Forschung und Entwicklung(IKFE) Berlin GmbH, Berlin
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - POLIKUM Institut GmbH, Berlin
  - DRK Kliniken Kopenick, Zentrum Klinische Forschung, Berlin
  - Berlin Research Centre-Synexus Clinical Research GmbH, Berlin
  - Synexus Clinical Research GmbH, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Medizinisches Versorgungszentrum am Bahnhof Spandau, Berlin
  - Klinikum Bielefeld, Bielefeld
  - Bochum Research Centre-Synexus Clinical Research GmbH, Bochum
  - MediClin Reha-Zentrum Spreewald, Burg
  - Klinikum Coburg, Coburg
  - Zentrum fuer klinische Forschung, Cologne
  - HELIOS Amper-Klinikum Dachau, Dachau
  - Kardiologische Praxisgemeinschaft, Dortmund
  - St. Johannes-Hospital, Dortmund
  - Gemeinschaftspraxis fuer Kardiologie Dres. Med. Willgeroth/Wetzel, Dortmund
  - Klinsche Forschung Dresden GmbH, Dresden
  - Praxis Dr. med. Christoph Axthelm, Dresden
  - GWT-TUD GmbH, Studienzentrum Professor Hanefeld, Dresden
  - Gemeinschaftspraxis Dr. Hagemann/Breiderhoff/Durfeld, Essen
  - Medizentrum Essen Borbeck, Essen
  - Studienzentrum, Essen
  - Gemeinschaftspraxis Dres. Dirk Weber, Ulrich Weber, Heiner Saueressig, Birte Turner und Georg, Essen
  - Schwerpunktpraxis Dr. Luedemann fuer Diabetes Gefaess- und Ernaehrungsmedizin, Falkensee
  - Clinphenomics Gmbh & Co Kg, Studienzentrum, Frankfurt
  - Synexus Clinical research GmbH, Frankfurt
  - IKF Institut fuer klinische Forschung Frankfurt, Frankfurt am Main
  - Klinik und Poliklinik fuer Innere Medizin B-Kardiologie, Angiologie, Pulmologie, Internistische, Greifswald
  - Cardiologicum Hamburg, Hamburg
  - Praxis Dr. med Cornelia Brauer, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Universitatsklinikum des Saarlandes Klinik fur Innere Medizin III, Homburgsaar
  - Praxis Dr. Heister, Kamp-Lintfort
  - Studienzentrum Dr. Appel, Kassel
  - Gemeinschaftspraxis Dr. Klein / Minnich, Künzing
  - Klinik fur Innere Medizin, Kardiologie und Angiologie MediClin Herzzentrum Lahr/Baden., Lahr
  - Synexus Clinical research GmbH, Leipzig
  - Synexus Leipzig Clinical Research Centre, Leipzig
  - Polikum Institut Leipzig GmbH, Leipzig
  - Gemeinschaftspraxis Dr. med. Heidrun Taeschner und Dr. med. Susanne Bonigut, Leipzig
  - Maerkische Kliniken GmbH, Klinikum Luedenscheid, Innere III, Lüdenscheid
  - Klinikum Lunen, St. Marienhospital, Lünen
  - SMO.MD GmbH - Zentrum fÃ¼r klinische Studien, Magdeburg
  - SMO.MD GmbH, Zentrum fuer klinische Studien Site Management and Clinical Research Unit, Magdeburg
  - Pfuetzner Science & Health Institute-Gmbh, Mainz
  - Staedtisches Klinikum Muenchen GmbH, Munich
  - Klinikum Der Universitat Munchen, München
  - Klinikum fuer Herz- & Kreislauferkrankungen, München
  - Kardiologische Praxis Northeim, Northeim
  - Gemeinschaftspraxis Drs Haggenmiller/Jeserich, Kardiologie, Angiologie, Innere Medizin, Nuremberg
  - Allgemeinmedizinisch-Internistische Praxisgemeinschaft, Offenbach
  - Praxis Dres. Med Naudts und Nowack, Rodgau
  - Klinik am See Rehabilitationszentrum fur Innere Medizin, Rüdersdorf
  - Kardiologische Gemeinschaftspraxis Dres Med. Gerke/Burger, Soest
  - Praxisgemeinschaft Stuhr-Brinkum, Stuhr-Brinkum
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Josephs-Hospital Warendorf Med. Klinik II, Kardiologie/Angiologie, Warendorf
  - Kardiologische Praxis, Wermsdorf
  - ForschungszentrumRuhr KliFoCenter GmbH, Witten
- Hungary (33):
  - Pecsi Tudomanyegyetem AOK, II., Pécs, Baranya
  - Bacs-Kiskun Megyei Korhaz, Kecskemét, Bács-Kiskun county
  - Szegedi Tudomanyegyetem AOK, I. sz Belgyogyaszati Klinika, Szeged, Csongrád megye
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár, Fejér
  - DRC Kft., Balatonfüred
  - DRC Kft., Balatongyörök
  - Grof Tisza Istvan Korhaz Berettyoujfalu, Berettyóújfalu
  - Kardiologiai Maganrendelo, Békéscsaba
  - Budapesti Szent Ferenc Korhaz, Budapest
  - Synexus Magyarorszag Kft, Budapest
  - Szent Rokus Korhaz, Budapest
  - Semmelweis Egyetem, Budapest
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Budapest
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz-Rendelointezet, Budapest
  - Egyesitett Szent Istvan Korhaz es Szent Laszlo Korhaz, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, III. Belgyogyaszat-Kardiologiai Osztaly, Budapest
  - Debreceni Egyetem, Debrecen
  - Synexus Magyarorszag Kft., Gyula
  - Edes Szivunk Egeszsegkozpont Kft., Hajdúszoboszló
  - BKS Research Kft., Albert Schweitzer Korhaz, Hatvan
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Jutrix Egeszsegugyi Kft, Kecskemét
  - Megyei Flor Ferenc Korhaz, Kistarcsa
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Josa Andras Oktatokorhaz, Nyíregyháza
  - Medifarma-98 Kft., Nyíregyháza
  - Pecsi Tudomanyegyetem AOK, I. Belgyogyaszati Klinika, Pécs
  - Mentahaz Maganorvosi Kozpont, Székesfehérvár
  - Hetenyi Geza Korhaz, Szolnok
  - Markusovszky Egyetemi Oktatokarhaz, Szombathely
  - Dr. Sydo es Tsa Kft., Veszprém
  - Zala Megyei Korhaz, Diabetológiai Szakrendelés, Zalaegerszeg
  - Zala Megyei Korhaz, Zalaegerszeg
- India (9):
  - Dr. Jivraj Mehta Smarak Health Foundation, Bakeri Medical Research Centre, Ahmedabad, Gujarat
  - Apex Heart Institute (A Unit of TCVS Pvt. Ltd), Ahmedabad, Gujarat
  - SAL Hospital, Ahmedabad, Gujarat
  - Apple Hospital, Surat, Gujarat
  - Unicare Heart Institute & Research Center, Surat, Gujarat
  - BAPS - Pramukh Swami Hospital, Surat, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
  - M.V. Hospital And Research Centre, Lucknow, Uttar Pradesh
- Ireland (2):
  - Beaumont Hospital, Dublin, Leinster
  - St James's Hospital, Dublin
- Israel (24):
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv
  - Barzilai Medical Center, Ashkelon
  - Ben Yair Community Clinic - Clalit Health Services, Beersheba
  - Heart Institute, Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - Cardiovascular Clinical Research Institute, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Cardiology Department, Nahariya
  - E.M.M.S Nazareth Hospital, Nazareth
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Rabin Medical Center-Beilinson Hospital, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Sha'aria Clinic, Clalit Health Services, Petah Tikva
  - Shuali Community Clinic, Clalit Health Services, Raanana
  - Department of Neurology & Sagol Neuroscience Center, Ramat Gan
  - Heart Institute, Kaplan Medical Center, Rehovot
  - Kaplan Medical Center Metabolism and Diabetes Clinic, Kaplan Medical Center, Rehovot
  - Internal Medicine A, Ziv Medical Center, Safed
  - Ziv Medical Center, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (22):
  - A.O. Treviglio e Caravaggio, Treviglio (BG), Bergamo
  - AOU Policlinico "Mater Domini" UOC di Medicina Interna, Catanzaro, CZ
  - Covance Central Laboratory Services, Meyrin/Geneve, Geneve
  - Ospedale S. L. Mandic di Merate, Merate, Lecco
  - Dipartimento delle Patologie Emergenti, Unita di Medicina Interna e Dislipidemie Genetiche, Palermo, PA
  - Ospedale S. Maria della Misericordia -Dipartimento di Medicina, Medicina Interna,, Perugia, PG
  - Azienda Ospedaliera Della Provincia Di Lecco - Ospedale Manzoni, Lecco, Province OF Lecco
  - Dip Medicina Interna e Specialita Mediche, Policlinico Umberto I, Roma, RM
  - Policlinico Umberto I di Roma, Rome, RM
  - Azienda Ospedaliera S'Andrea di Roma - UOC Cardiologia, Rome, RM
  - Ospedale G. Fracastoro, San Bonifacio, Verona
  - AOUI di Verona - Ospedale Civile Maggiore Borgo Trento, Verona, VR
  - S. C. Cardiologia INRCA, Ancona
  - Ospedale Civile Regionale San Martino, Belluno, Belluno
  - Azienda Ospedaliera G. Brotzu, Cagliari
  - Unità Operativa Solventi e Unità Poliambulatorio, Milan
  - Department of Clinical Medicines and Cardiovascular Sciences, Universita "Federico II" di Napoli, Napoli
  - Divisione di Cardiologia con Utic ed Emodinamica - AOU Federico II di Napoli, Napoli
  - A.O. di Reggio Emilia Arcispedale "S. Maria Nuova"/IRCCS, Reggio Emilia
  - AUSL Della Romagna-Ospedale Infermi, Rimini
  - Ospedale Santa Maria della Misericordia Azienda ULSS 18 of Rovigo, Rovigo
  - Azienda Ospedaliera Universitaria Santa Maria della Misericordia, Udine
- Mexico (37):
  - Consultorio Dr. Leocadio Gerardo Munoz Beltran, Cd. Juarez, Chihuahua
  - Centro de Investigacion Clinica del Pacifico, S.A. de C.V., Acapulco de Juárez, Guerrero
  - Hospital Del Pacifico,Centro De Investigacion Clinica Del Pacifico Cicpa,Torre Medica Del Pacifico, Acapulco de Juárez, Guerrero
  - Clinical Trials Mexico, S.A. de C.V., Pachuca, Hidalgo
  - Investigacion Biomedica Aplicada de Hidalgo S.A. de C.V., Pachuca, Hidalgo
  - Centro de Investigacion Medica Integral S.C., Guadalajara, Jalisco
  - Icle S.C., Guadalajara, Jalisco
  - Consultorio Privado del Dr. Gabriel Arturo Ramos Lopez, Guadalajara, Jalisco
  - Unidad de Investigacion Clinica y Atencion Medica Hepa S.C., Guadalajara, Jalisco
  - Consultorio de Endocrinologia y Nutriologia, Mexico City, Mexico City
  - Operadora de Hospitales Angeles S.A. de C.V. (Emergencies), Mexico City, Mexico City
  - Centro Especializado en Diabetes Obesidad y Prevencion de Enfermedades Cardiovasculares, SC., Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion "Salvador Zubiran", Mexico City, Mexico City
  - Instituto de Diabetes Obesidad y Nutricion, S.C., Cuernavaca, Morelos
  - Hospital Inovamed Cuernavaca (Emergencies), Cuernavaca, Morelos
  - Cardiolink Clin Trials, S.C., Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - CRI Centro Regiomontano de Investigacion SC, Monterrey, Nuevo León
  - Global Trial Research Center S.A. de C.V., Monterrey, Nuevo León
  - Centro Integral Medico SJR S.C, San Juan del Río, Querétaro
  - Centro para el Desarrollo de la Medicina y de Asistencia Médica Especializada S.C., Culiacán, Sinaloa
  - Hospital Angeles Culiacan, Culiacán, Sinaloa
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares S.C., Tampico, Tamaulipas
  - Centro De Especialidades Medicas Del Estado De Veracruz, Xalapa, Veracruz
  - Instituto Biomedico De Investigacion A.C., Aguascalientes
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Unidad De Investigacion En Salud De Chihuahua S.C., Chihuahua City
  - Consultorio Medico de Especialidad Dr. Demetrio Kosturakis Garcia, Chihuahua City
  - Investigacion en Salud y Metabolismo S.C, Chihuahua City
  - Instituto Nacional de Ciencia Medicas y Nutricion Salvador Zubiran, Distrito Federal
  - Lahoja Asociacion para la Investigacion y Farmacovigilancia S.C., Durango
  - Centro Especializado en Diabetes, Obesidad y Prevencion de Enfermedades Cardiovasculares, S.C., México
  - Pharmacology and Clinical Research S.A. de C.V., Querétaro
  - Cardioarritmias e Investigacion S.C., San Luis Potosí City
  - Hospital Lomas de San Luis lntemacional (Emergencies), San Luis Potosí City
  - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City
  - Centro Especializado En Diabetes Y Metabolismo, Veracruz
- Netherlands (74):
  - Zuyderland MC, Sittard-Geleen, Limburg
  - Isala, Zwolle, Overijssel
  - Tjongerschans Ziekenhuis, Heerenveen, Provincie Friesland
  - St. Franciscus Gasthuis, Rotterdam, South Holland
  - Het Lange Land Ziekenhuis, Zoetermeer, South Holland
  - Noordwest Ziekenhuisgroep, Alkmaar
  - EB Flevoresearch, Almere Stad
  - Meander Medical Center, Amersfoort
  - Meander Medisch Centrum, Amersfoort
  - Amstelland Hospital, Amstelveen
  - Bovenij Ziekenhuis, Amsterdam
  - OLVG, locatie West, Amsterdam
  - VU University Medical Center, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academic Medical Center, Amsterdam
  - Gelre Hospitals, Apeldoorn
  - Rode Kruis Ziekenhuis, Beverwijk
  - Tergooi Ziekenhuis, Blaricum
  - Andro Medical Research B.V., Breda
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Ziekenhuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Van Weel Bethesda Hospital, Dirksland
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer Ziekenhuis-Albert Schweitzer Hospital, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Andromed Eindhoven, Eindhoven
  - Heartcentre Catharina Hospital, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Beatrix Hospital, Gorinchem
  - Beatrix Ziekenhuis, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - University Medical Center Groningen, Groningen
  - Martini Ziekenhuis, Groningen
  - Spaarne Gasthuis, Haarlem
  - Ropcke Zweers Hospital, Hardenberg
  - St. Jansdal Ziekenhuis, Harderwijk
  - Zuyderland Medisch Centrum, Heerlen
  - Zuyderland, Heerlen
  - Treant Zorggroep, location Bethesda, Hoogeveen
  - Vascular Research Centre, Hoorn
  - Quality Care Research, Kloosterhaar
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Alrijne Ziekenhuis, Leiden
  - Alrijne Ziekenhuis, Leiderdorp
  - GCM Maarssenbroek, Maarssen
  - Maastricht University Medical Center, Maastricht
  - Isala Diaconessenhuis, Meppel
  - St Antonius Hospital, Nieuwegein
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Waterland Hospital, Purmerend
  - Andro Medical Research B.V., Rotterdam
  - Hedramed, Rotterdam
  - Rotterdam Research Institute, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - D&A Research and Genetics, Sneek
  - Hedramed, The Hague
  - Hagaziekenhuis, The Hague
  - Bronovo Ziekenhuis, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Elisabeth-TweeSteden Ziekenhuis (previously named St. Elisabeth Ziekenhuis), Tilburg
  - St. Elisabeth Ziekenhuis, Tilburg
  - Elisabeth TweeSteden Ziekenhuis (ETZ), Tilburg
  - Bernhoven Ziekenhuis, Uden
  - EB Utrecht, Utrecht
  - Universitair Medisch Centrum (UMC) Utrecht - Locatie AZU, Utrecht
  - University Medical Center Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - VieCuri Medisch Centrum, Venlo
  - Twee Steden Ziekenhuis, Waalwijk
  - Klinisch Onderzoek Praktijk Zoetermeer, Zoetermeer
  - Albert Schweitzer Hospital, Zwijndrecht
- New Zealand (19):
  - Henderson Medical Centre, Henderson, Auckland
  - North Shore Hospital, Takapuna, Auckland
  - Hawke's Bay Hospital, Frimley, Hastings
  - North Shore Hospital, Laboratory, Auckland
  - North Shore Hospital- Inpatient Pharmacy, Auckland
  - Optimal Clinical Trials, Auckland
  - Auckland City Hospital, Auckland
  - Middlemore Clinical Trials, Auckland
  - Lipid and Diabetes Research Group, Christchurch
  - Southern Clinical Trials Shirley Ltd Don Beavan Medical Research Centre, Christchurch
  - Southern Clinical Trials Riccarton, Christchurch
  - Taranaki Base Hospital, New Plymouth
  - Papamoa Pines Medical Centre, Papamoa
  - Rotorua Hospital, Rotorua
  - Clinical Horizons NZ Ltd, Tauranga
  - Clinical Trials Unit,Bay of Plenty(BOP) Clinical School, Tauranga
  - CCDHB, Wellington Hospital, Clinical Measurement Unit, Wellington
  - Wellington Hospital, Wellington
  - Wellington Regional Hospital, Wellington
- Poland (83):
  - Synexus Polska Sp. z o.o Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Nzoz "Twoja Przychodnia", Poznan, Greater Poland Voivodeship
  - SPZOZ Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej Uniwersytetu Medycznego, Lodz, Iodzkie
  - NZOZ Vitamed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Nzoz Centrum Medyczne Kermed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczna Praktyka Lekarska Piotr Kubalski, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczne Gabinety Lekarskie "Medicor Plus" - Jerzy Kopaczewski, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Landa Specjalistyczne Gabinety Lekarskie, Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. J. Dietla w Krakowie, Oddzial Kardiologii, Krakow, Lesser Poland Voivodeship
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Oddzial Szybkiej Diagnostyki, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Zdrowa J. Trebacz, W. Zajdel Spolka Jawna, Krakow, Lesser Poland Voivodeship
  - CENTRUM MEDYCZNE A-Z Clinic, Krakow, Lesser Poland Voivodeship
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki W Krakowie,, Krakow, Lesser Poland Voivodeship
  - NeuroCor Banaszkiewicz, Kulaga, Ostrowska, Tomaszewski lekarze spolka partnerska, Myślenice, Lesser Poland Voivodeship
  - INTERCARD Sp. z. o. o. Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii w Nowym Targu, Nowy Targ, Lesser Poland Voivodeship
  - Centrum Szybkiej Diagnostyki Kardiologicznej Kardiomed M. Zabowka E. Zabowka, Tarnów, Lesser Poland Voivodeship
  - Specjalistyczny Gabinet Lekarski Internistyczno-Kardiologiczny Boguslaw Derlaga, Tarnów, Lesser Poland Voivodeship
  - Jeleniogorskie Centrum Chorob Serca, Przychodnia Kardiologiczna, Poradnia Kardiologiczna, Jelenia Góra, Lower Silesian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Osrodek Badawczo-Rozwojowy, Wroclaw, Lower Silesian Voivodeship
  - Zdrowie s.c. Agnieszka i Donald Drozdz, Wroclaw, Lower Silesian Voivodeship
  - Halina Serafin NZOZ Centrum Medyczne SERAFIN-MED, Żarów, Lower Silesian Voivodeship
  - Clinical Best Solutions, Lublin, Lublin Voivodeship
  - Optimamed Specjalistyczne Gabinety Lekarskie, Lublin, Lublin Voivodeship
  - KO-MED Centra Kliniczne Lublin II, Lublin, Lublin Voivodeship
  - KO-MED Centra Kliniczne Pulawy, Puławy, Lublin Voivodeship
  - KO-MED Centra Kliniczne Zamosc, Zamość, Lublin Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Masovian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Specjalistyczna Przychodnia Lekarska "MEDIKARD", Płock, Masovian Voivodeship
  - Centrum Medyczne Piaski Filia Nr 9, Warsaw, Masovian Voivodeship
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych w Warszawie, Warsaw, Masovian Voivodeship
  - CSK MSW w Warszawie, Klinika Kardiologii Zachowawczej i Nadcisnienia Tetniczego, Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny, Klinika Kardiologii i Chorob Wewnetrznych, Centralny Szpital Kliniczny, Warsaw, Masovian Voivodeship
  - Instytut Kardiologii im. Prymasa Tysiaclecia Stefana Kardynala Wyszynskiego, Warsaw, Masovian Voivodeship
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego Sp. z o.o., Warsaw, Masovian Voivodeship
  - Szpital Specjalistyczny w Brzozowie, Podkarpacki Osrodek Onkologiczny im. Ks. B. Markiewicza Oddzial, Brzozów, Podkarpackie Voivodeship
  - INTERCARD Sp. z o.o. Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii w Krosnie, Krosno, Podkarpackie Voivodeship
  - EMED Centrum Uslug Medycznych Ewa Smialek, Rzeszów, Podkarpackie Voivodeship
  - """OSTEO-MEDIC"" s.c. Artur Racewicz, Jerzy Supronik", Bialystok, Podlaskie Voivodeship
  - Podlaski Osrodek Kardiologii Janusz Korecki, Bialystok, Podlaskie Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk, Pomeranian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Gdanskie Centrum Zdrowia, Poradnia Kardiologiczna, Gdansk, Pomeranian Voivodeship
  - Centrum Badan Klinicznych Pi-House, Poradnia Diabetologiczna, Gdansk, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - NZOZ "PRO CORDIS" Sopockie Centrum Badan Kardiologicznych, Gdynia, Pomeranian Voivodeship
  - Gabinet Kardiologiczno - lnternistyczny, Gdynia, Pomeranian Voivodeship
  - Centrum Medyczne "SOPMED" Sp. z o.o., Sopot, Pomeranian Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska Malgorzata Biedrzycka, Starogard Gdański, Pomeranian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Wojewodzki Szpital Specjalistyczny Nr 4 w Bytomiu,, Bytom, Silesian Voivodeship
  - Bogna Gabrylewicz Andrzej Ochala Unimed s.c., Katowice, Silesian Voivodeship
  - Pro Familia Altera Poradnia Wielospecjalistyczna, Katowice, Silesian Voivodeship
  - NZOZ Terapia Optima, Katowice, Silesian Voivodeship
  - Przychodnia Specjalistyczna Samodzielny Publiczny ZOZ w Rudzie Slaskiej, Poradnie Specjalistyczne,, Ruda Śląska, Silesian Voivodeship
  - NZOZ "Medyk"Sp. z o. o., Wola, Silesian Voivodeship
  - Wojewodzki Szpital Zespolony w Elblagu, Oddzial Kardiologiczny z Pododdzialem Kardiologii Inwazyjnej, Elblag, Warmian-Masurian Voivodeship
  - "OSTEO-MEDIC" s.c. Artur Racewicz, Jerzy Supronik, Bialystok
  - NZOZ Vitamed -Ga¿aj I Cichomski sp.j, Bydgoszcz
  - Medica Pro Familia Sp. z o.o. Spolka Komandytowo Akcyjna, Oddzial w Gdyni, Gdynia
  - Nzoz Gall-Med, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie,, Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - NZOZ Centrum Zdrowia i Profilaktyki Dabie Sp. z.o.o., Krakow
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego, Lodz
  - "TWOJA PRZYCHODNIA" Sp. Z o.o, Lublin
  - NeuroCor Banaszkiewicz, Kulaga, Ostrowska, Tomaszewski lekarze spolka partnerska, Myślenice
  - Medicus w Opolu Sp z o. o., Opole
  - Specjalistyczny Osrodek Leczniczo-Badawczy Zbigniew Zegota, Ostróda
  - Medicome Sp. z o.o., Oświęcim
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - NZOZ Przychodnia Specjalistyczna Andrzej wittek Henryk Rudzki S.C., Ruda Śląska
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Instytut Kardiologii, Ii Klinika Choroby WieCowej, Warsaw
  - Instytut Kardiologii im. Prymasa Tysiaclecia Stefana Kardynala Wyszynskiego, Warsaw
  - Instytut Kardiologii im. Prymasa Tysiaclecia Stefana Kardynala, Warsaw
  - Dobrostan Michal Bogacki, Wroclaw
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz, Łódź Voivodeship
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego Sp. z o.o., Lodz, Łódź Voivodeship
  - "Prywatny Gabinet Kardiologiczny" Dr N.Med. Maciej Kosmider, Lodz, Łódź Voivodeship
  - Prywatny Gabinet Lekarski Dr n. med. Michal Ogorek, Piotrkow Trybunalski, Łódź Voivodeship
  - Centrum Medyczne Ogrodowa Sp. z o.o., Skierniewice, Łódź Voivodeship
  - Prywatny Gabinet Lekarski Marianna Janion, Kielce, Świętokrzyskie Voivodeship
- Puerto Rico (7):
  - Cardiometabolic Research Center, Inc., Ponce, PR
  - Endocrine Lipid Diabetes Research Institute, Ponce, PR
  - Miguel Sosa-Padilla, MD-Private Practice, San Juan, PR
  - The Office of Roberto J. Ayala-Rios, MD - Research Center and Private Practice (DMRA LLC), Añasco
  - Pradnet Inc., San Juan
  - Altamira Family Medicine And Research Institute, San Juan
  - Centro de Diabetes para Puerto Rico, San Juan
- Romania (34):
  - Pitesti-Arges County Emergency Hospital, Piteşti, Argeş
  - Medical Practice SRL, Oradea, Bihor County
  - County Clinical Emergency Hospital Oradea, Oradea, Bihor County
  - County Emergency Hospital Deva, Deva, Hunedoara County
  - CMI Pop Calin Florin, Baia Mare, JUD Maramures
  - Centrul Medical Dr. Negrisanu SRL, Diabet Zaharat Nutritie si Boli Metabolice, Timișoara, Judet Timis
  - Dr. Pop Calin Florin - Cabinet Cardiologie, Baia Mare, Maramureş
  - Podoleanu G. Cristian-Gheorghe-Calin - Cardiology Medical Practice, Târgu Mureş, Mureș County
  - Diabmed Dr. Popescu Alexandrina SRL, Diabet, Nutritie, Boli Metabolice, Ploieşti, Prahova
  - Dr. Busegeanu Mihaela Private Practice, Ploieşti, Prahova
  - Clinica Medicala Synexus Ltd., Bucharest, Sectorul 2
  - Institute of Cardiovascular Diseases Timisoara, Timișoara, Timiș County
  - Euromedica Hospital, Baia Mare
  - S.C. Polimed Dacia S.R.L., Brasov
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL, Medicina Interna, Brasov
  - Spitalul Clinic Judetean De Urgenta Braila(Braila County Clincal Emergency Hospital), Brăila
  - Data Plus Medical Clinic, Bucharest
  - Spitalul Universitar De Urgenta Militar Central, Dr. Carol Davila, Bucharest
  - "Prof. Dr. N.C. Paulescu" National Institute of Diabetes, Nutrition and Metabolic Diseases,, Bucharest
  - Spitalul Clinic Colentina, Departament Cardiologie, Bucharest
  - SC Centrul Medical Policlinico Di Monza SRL, Cardiologie, Bucharest
  - SC Policlinica CCBR SRL, Bucharest
  - Med Plus SRL (Med Plus Ltd.), Bucharest
  - S.C. Centrul Medical "Sanatatea Ta" S.R.L., Bucharest
  - Med Plus Srl, Bucharest
  - Spitalul Clinic Judetean De Urgenta Cluj-Napoca, Diabet Zabarat, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Diabet Zaharat, Nutritie si Boli Metabolice, Cluj-Napoca
  - Dr. Mistodie Cristina Victoria MD, Office of, Galati
  - S.C. Diamed Obesity S.R.L., Galati
  - County Emergency Hospital Satu Mare Diabetes, Nutrition And Metabolic Diseases Department, Satu Mare
  - County Clinical Emergency Hospital Sibiu, Sibiu
  - Cardio Med SRL, Cardiologie, Tg. Mures
  - Centrul Medical Sf. Stefan, Timișoara
  - Institution Centrul Medical Sf. Stefan SRL, Diabet Nutritie si Boli Metabolice, Timișoara
- Russia (61):
  - State Budgetary Healthcare Institution "Research Institution - Regional Clinical Hospital #1, Krasnodar, Krasnodarskiy Kray
  - State Budgetary Healthcare Institution of Moscow Region "Lubertsy Regional Hospital #2", Lubertsy, Moscow Oblast
  - Federal State Budgetary Institution of Healthcare Hospital of Russian Academy of Sciences, Troitsk, Moscow Oblast
  - 1st Pavlov State Medical University of St. Petersburg, Saint Petersburg, Sankt-Peterburg
  - Saint Petersburg State Budgetary Institution of Healthcare, Saint Petersburg, Sestroretsk
  - FSBEI of HE Kazan State Medical University on the base of SBHI Clinical Hospital No.2, Kazan', Tatarstan Republic
  - Municipal Budgetary State Healthcare Institution "City Clinical Hospital #6", Chelyabinsk
  - Non-State Institution of Healthcare, Chelyabinsk
  - State Budgetary Healthcare Institution ¿Region Clinical Hospital #3¿, Chelyabinsk
  - Regional Budgetary Healthcare Institution "Cardiology Dispensary", Ivanovo
  - State Budgetary Institution of Healthcare of Kaluga Region "Kaluga Regional Hospital", Kaluga
  - Federal State Budgetary Educational Institution of Higher Education "Kazan State Medical University", Kazan'
  - State Autonomous Healthcare Institution "Republic Clinical Hospital", Kazan'
  - "SAHI of Kemerovo ""Regional Clinical Hospital of Emergency Medical Care n.a. M.A Podgorbunsky """, Kemerovo
  - Municipal Budgetary Institution of Healthcare Municipal Clinical Hospital #3 n.a. M.A. Podgorbunsky, Kemerovo
  - FSBI "Research institute of complex problems of cardio-vascular diseases" of, Kemerovo
  - FSHI "Medical and Sanitary Unit of the Ministry of Internal Affairs of Russia across, Kemerovo
  - Kirov Regional State Budgetary Healthcare Institution "Kirov City Clinical Hospital #1", Kirov
  - Regional Budgetary Healthcare Institution "Kursk City Clinical Emergency Hospital", Kursk
  - Non-State Institution of Healthcare "Central Clinical Hospital #6 OAO "RZhD", Moscow
  - SBHI Moscow city "City Clinical Hospital #15 n.a. O.M. Filatova" of Moscow Healthcare Department, Moscow
  - Federal State Budgetary Institution "Central Clinical Hospital with Polyclinic", Moscow
  - "Federal State Budgetary Institution "Russian Cardiology Research And Production Complex" Of, Moscow
  - Moscow State Healthcare Institution "City clinical hospital n.a. S.P.Botkin", Moscow
  - State Budget Institution of Healthcare (SBIH) of Moscow "City Clinical Hospital #81, Moscow
  - Federal State Budget Institution "Out-patient Clinic #3" of Russian Federation, President's, Moscow
  - State Regional Budgetary Healthcare Institution, Murmansk
  - State Budgetary Healthcare Institution of Nizhegorodskaya Region, Nizhny Novgorod
  - Federal State Budgetary Institution "Research Institute of Therapy and Preventive Medicine", Novosibirsk
  - "Reafan" LLC, Novosibirsk
  - Municipal Budgetary Institution of Healthcare of Novosibirsk, Novosibirsk
  - State Budgetary Institution of Healthcare of Novosibirsk region City Clinical Hospital of Emergency, Novosibirsk
  - State Budgetary Healthcare Institution (SBHI) N.N. Burdenko Regional Clinical Hospital of Penza, Penza
  - SBHI of Saint-Petersburg "City Hospital # 38 n.a. N.A. Semashko", Pushkin
  - State Budgetary Educational Institution Of Higher Professional Education, Rostov-on-Don
  - State Budgetary Educational Institution of Higher Professional Education, Rostov-on-Don
  - State Budgetary Institution "Ryazan Regional Clinical Hospital", Ryazan
  - Saint-Petersburg State Budgetary Institution of Healthcare "City Hospital #23", Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City Alexandrovskaya Hospital", Saint Petersburg
  - Limited Liability Company "Reavita", Saint Petersburg
  - LLC "Institution of medical studies", Saint Petersburg
  - Saint-Petersburg State Budgetary Institution of Healthcare "City Hospital #26", Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Academician I.P. Pavlov First, Saint Petersburg
  - SBEI of HPE "First Pavlov State Medical University of St. Petersburg" of the MoH of the RF, Saint Petersburg
  - Federal State Budgetary Institution "Advisory Diagnostic Center and Polyclinic", Saint Petersburg
  - Federal State Budgetary Institution "Federal Almazov Medical Research Centre" of, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City Hospital #15", Saint Petersburg
  - Limited Liability Company International Medical Centre SOGAZ, Saint-Petersberg
  - State Budgetary Healthcare Institution "Samara Regional Clinical Cardiology Dispensary", Samara
  - MHI "City Clinical Hospital 12"of the Healthcare Committee of, Saratov
  - State Institution of Healthcare "Regional Clinical Hospital", Saratov
  - Tyumen Cardiology Research Center-branch of the Tomsk NRMC, Tomsk
  - State Budgetary Educational Institution of Highest Professional Education, Tomsk
  - State Autonomous Healthcare Institution of Tyumen region "Scientific-Practical Medical Center", Tyumen
  - "Tyumen Cardiology Center" Affiliate of the FSBSI "Scientific and Research Institution of Cardiology, Tyumen
  - State Autonomous Healthcare Institution of Yaroslavl region Clinical Emergency Hospital n.a..N.V.So, Yaroslavl
  - State Autonomous Healthcare Institution of Yaroslavl Region, Yaroslavl
  - FSBEI of HE "Yaroslavl State Medical University" MH of the Russian Federation based on Clinical, Yaroslavl
  - State Budgetary Healthcare Institution of Yaroslavl Region "Clinical Hospital No. 10", Yaroslavl
  - State Healthcare Institution of Yaroslavl Region "Clinical Hospital #8", Yaroslavl
  - Municipal Autonomous Institution "City Clinical Hospital #14", Yekaterinburg
- Slovakia (41):
  - Nemocnica Ruzinov-Univerzitna Nemocnica Bratislava (UNB), Bratislava, Bratislava Region
  - Stredoslovensky ustav srdcovych a cievnych chorob a.s., Banská Bystrica
  - Fakultna nemocnica F. D. Roosevelta, Banská Bystrica
  - Alian s.r.o., kardiologicka ambulancia, Bardejov
  - Metabol KLINIK s.r.o., Ambulancia pre diabetologiu, poruchy latkovej premeny a vyzivy, Bratislava
  - Univerzitna nemocnica Bmtislava, Nemocnica Stare Mesto, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Stare Mesto, l.interna klinika, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Stare Mesto, Bratislava
  - UN Bratislava, Nemocnica Ruzinov, V. interna klinika LFUK a UN Bratislava, Bratislava
  - Kardiovaskularne Centrum S.R.O., Bratislava
  - Metabolicke Centrum MUDr. Katariny Raslovej, S.R.O., Bratislava
  - Narodny ustav srdcovych a cievnych chorob, a.s., Bratislava
  - Univerzitna Nemocnica Bratislava, Bratislava
  - KARDIO-SANUS spol.,s.r.o.,Kardiologicka, interna a sonograficka ambulancia, Bratislava
  - KARDIO-SANUS spol. s.r.o., Bratislava
  - VERIA, s.r.o. -Kardiologicka ambulancia, Bratislava
  - UN Bratislava Nemocnica Sv.Cyrila a Metoda, kardiologicka ambulancia 1, Bratislava
  - Endiamed s.r.o. Nestatna diabetologicka a endokrinologicka ambulancia, Dolný Kubín
  - JM-Interna s.r.o., interna ambulancia, Dolný Kubín
  - CARDIO D&R s.r.o., Kardiologicka ambulancia, Košice
  - AGTO., spol. s r. o., Košice
  - Cardio D&R spol.s.r.o., kardiologicka ambulancia, Košice
  - Medicentrum Heart, Spol. S.R.O, Kráľovský Chlmec
  - CELL-B s.r.o. interna ambulancia, Levice
  - Liptovska nemocnica s poliklinikou MUDr.Ivana Stodolu Liptovsky Mikulas, Liptovský Mikuláš
  - KARDIO 1 s.r.o., Lučenec
  - Narodny Endokrinologicky A Diabetologicky Ustav N.O., Ľubochňa
  - Klinika hematologie a transfuziologie, Univerzitna nemocnica Martin, Martin
  - MEDI M&M s.r.o., Ambulancia vnutorneho lekarstva, Moldava nad Bodvou
  - MUDr. Kanderkova s.r.o., Diabetologicka ambulancia, Námestovo
  - Kardiocentrum Nitra s.r.o., kardiologicka ambulancia, Nitra
  - Fakultna nemocnica s poliklinikou Nove Zamky, I. interna klinika, Nové Zámky
  - Mediab s.r.o. Diabetologicka ambulancia, Pezinok
  - BENIMED s.r.o., Piešťany
  - Medispol S.R.O., Prešov
  - Medilex s.r.o. Interna ambulancia, Rimavská Sobota
  - Kardioamb S.R.O., Rimavská Sobota
  - DIAMEL, s.r.o., Diabetologicka ambulancia, Trenčín
  - BV Medical, s.r.o. Diabetologicka ambulancia,, Trnava
  - Kardiologicka ambulancia, Trnava
  - Medivasa S.R.O., Diabetologicka Ambulancia, Žilina
- South Africa (31):
  - IATROS International, Bloemfontein, Free State
  - JOSHA Research, Bloemfontein, Free State
  - Welkom Clinical Trial Centre, Welkom, Free State
  - Midrand Medical Centre, Halfway House, Gauteng
  - Centre for Diabetes and Endocrinology, Houghton Estate, Gauteng
  - Sunninghill Hospital, Johannesburg, Gauteng
  - I Engelbrecht Research (Pty) Ltd, Lyttelton, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Gauteng
  - Medipark Centre for Clinical Research, Pretoria, Gauteng
  - Synexus Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Jongaie Research, Pretoria West, Gauteng
  - Roodepoort Medicross Clinical Research Centre, Roodepoort, Gauteng
  - Wits Clinical Research-Chris Hani Baragwanath Hospital, Soweto, Gauteng
  - Medi-Clinic Heart Hospital, Sunnyside, Gauteng
  - Suite 502, Durban, KwaZulu-Natal
  - Dr Ganesh c/o Dr NB Maharaj, Durban, KwaZulu-Natal
  - Nash Ranjith Research Centre, Merebank, Durban, KwaZulu-Natal
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - Zinakekele Medical Centre, Moloto South, Mpumalanga
  - Drs Joynt Venter & Associates, Witbank (eMalahleni), Mpumalanga
  - Dr JM Engelbrecht Trial Site-Vergelegen Mediclinic, Cape Town, Western Cape
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Synopsis Research cc, Cape Town, Western Cape
  - Helderberg Research Institute, Somerset West, Western Cape
  - Synexus Helderberg Clinical Research Centre, Somerset West, Western Cape
  - Vergelegen Mediclinic-Helderberg Research Institute, Somerset West, Western Cape
  - Unitas Hospital., Centurion
  - Clinresco Centres (Pty) Ltd-Central Professional Suits, Gauteng
  - Paarl Research Centre, Paarl
  - TREAD Research cc, Parow
  - Clinical Projects Research SA (Pty) Ltd, Worcester
- South Korea (21):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheonbuk-do
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Yonsei University Wonju College of Medicine, Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Uijeongbu St. Mary's Hospital-The Catholic University of Korea, Uijeongbu-si, Gyeonggi-do
  - Donguk University Gyeongju Hospital, Gyeongju, Gyeongsangbuk-do
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University Of Korea Seoul St.Marys Hospital, Seoul
  - Seoul Metropolitan Government - Seoul National University Boramae Medical Center, Seoul
- Spain (67):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Virgen De Los Lirios, Alcoy, Alicante
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Comarcal d'Inca, Inca, Balearic Islands
  - Cap Florida, L'Hospitalet de Llobregat, Barcelona-cataluna
  - CAP Disset De Setembre (Sant Cosme I Sant Damia), el Prat de Llobregat, Barcelona/cataluna
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - CAP La Mina, Sant Adrià de Besòs, Barcelona
  - EAP Vic, Vic, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Basque Country
  - Hospital Universitario Marques De Valdecilla, Santander, Cantabria
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona, Catalonia
  - Albera Salut, Peralada, Gerona
  - Hospital De Figueres, Figueres, Girona-catalonia
  - Hospital Santa Caterina, Salt, Girona, Girona
  - Hospital Arquitecto Marcide, Ferrol, LA Coruna
  - Hospital Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Centro de Salud El Cristo, Oviedo, Principality of Asturias
  - Centro Salud Paulino Prieto, Oviedo, Principality of Asturias
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitario San Juan de Alicante, Alicante, Valencia
  - Hospital General De Requena, Requena, Valencia
  - Gerencia de Gestion integrada de A Coruna, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante; Servicio Cardiologia, Alicante
  - Hospital Virgen del Mar, Almería
  - Parc de Salut mar ¿ Hospital del Mar, Barcelona
  - Parc de Salut Mar- Hospital del Mar, Barcelona
  - Centre Teknon, Barcelona
  - EAP Sardenya, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - CAP Centelles, Barcelona
  - CAP Amadeu Torner, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Fundacio Hospital de I'Esperit Sant, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Complexo Hospitalario Universitario Arquitecto Marcide-Profesor Novoa Santos De Ferrol, Ferrol
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves (HUVN), Granada
  - Hospital Universitari Arnau de Vilanova (HUAV), Lleida
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Pharmacy - Hospital Universitari Arnau de Vilanova (HUAV), Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Carlos III, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz; Unidad Metabolico-Vascular, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Carretera Alcala-Meco s/n, Madrid
  - H. U. Principe de Asturias, Madrid
  - Hospital Universitario Virgen de la Victoria. CE San Jose Obrero, Málaga
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Sant Joan de Reus, Reus (Tarragona)
  - Clinica Nuevas Tecnologias En Diabetes Y Endocrinologia, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - CAP Muralles, Tarragona
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clinico Universitario Miguel Servet; Medicina Interna, Zaragoza
- Sweden (18):
  - Karolinska universitetssjukhuset Huddinge, Stockholm, Huddinge
  - Kasernens Läkarservice AB, Eksjö
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Pharmasite AB, Helsingborg
  - Medicinklinikens forskningsenhet, Kristianstad
  - Hjartmottagningen, Capio Citykliniken, Lund
  - Probar E Lund AB, Lund
  - Karlkliniken, Skanes Universitetssjukhus i Malmo, Malmo
  - Pharmasite AB, Malmo
  - Forskningsenheten, Medicinmottagningen Sahlgrenska Universitetssjukhuset/Molndal, Hus J, Mölndal
  - Ostersunds Sjukhus, Östersund
  - Dalecarlia Clinical Research Center, Rättvik
  - Skelleftea Lasarett, Skellefteå
  - A+Science City site, Stockholm
  - Karolinska Universitetssjukhuset, Stockholm
  - Hjartkliniken, Stockholm
  - Akademiska Sjukhuset, Uppsala
  - Vastmanlands Sjukhus Vasteras, Västerås
- Switzerland (10):
  - Diagene Laboratories Inc., Reinach, Basel
  - Universitatsspital, Basel, Canton of Basel-City
  - Hospitaux Universitaires de Geneve (HUG), Geneva, Canton of Geneva
  - Policlinique Medicale Universitaire, Lausanne, Canton of Vaud
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Luzerner Kantonsspital Luzern, Lucerne
  - Cardiocentro Ticino, Lugano
  - Fondazione Diabete Lugano, Lugano
  - Kantonsspital St. Gallen, Sankt Gallen
- Taiwan (9):
  - China Medical University Hospital, Taichung, Taiwan R O C
  - National Taiwan University Hospital, Taipei, Taiwan R O C
  - Kaohsiung Medical University Chung-Ho Memorial Hospital - New, Kaohsiung City
  - Cardinal Tien Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University (NCKU) Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (5):
  - Division of Cardiology, Department of Medicine, Faculty of Medicine, Siriraj Hospital,, Bangkoknoi, Bangkok
  - Faculty of Medicine, Srinagarind Hospital, Khon Kaen University, Muang, Changwat Khon Kaen
  - Heart Center, Songklanagarind Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Cardiology Unit,Department of Medicine, Faculty of Medicine, Ramathibodi Hospital,, Bangkok
  - Division Of cardiology,Department of Medicine,Faculty Of Medicine,Chulalongkorn University, Bangkok
- Turkey (Türkiye) (20):
  - Baskent University, Adana Yuregir Training & Research Hospital, Adana
  - A.karahisar Kocatepe Universitesi Hastanesi Ahmet Needet Sezer Uygulama ve, Afyonkarahisar
  - Diskapi Yildirim Beyazit Egitim ve Arastirma Hastanesi, Ankara
  - Ufuk University School of Medicine, Dr. Ridvan Ege Training & Research Hospital, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Antalya Training & Research Hospital, Antalya
  - Adnan Menderes Universitesi Uygulama ve Arastirma Hastanesi, Aydin
  - Bursa Yuksek Ihtisas Egitim ve Arastirma Hastanesi, Bursa
  - Firat Universitesi, Elâzığ
  - Gaziantep Universitesi Tip Fakultesi Sahinbey Egitim ve Arastirma Hastanesi, Gaziantep
  - Bezmialem Vakif Universitesi Tip Fakultesi Kardiyoloji Bolurnu, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Istanbul Universitesi Kardiyoloji Enstitusu, Istanbul
  - Ege University, School of Medicine, Izmir
  - Izmir Tepecik Egitim ve Arastirma Hastanesi, Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi Hastanesi, Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Kocaeli University School Of Medicine-Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Mersin University, School of Medicine, Mersin
  - Recep Tayyip Erdogan University School of Medicine, Training & Research Hospital, Rize
- United Kingdom (49):
  - Synexus Thames Valley Clinical Research Centre, Reading, Berkshire
  - Peterborough and Stamford Hospitals NHS Foundation Trust, Peterborough, Cambridgeshire
  - Brannel Surgery, St Austell, Cornwall
  - Queens Hospital, Romford, Essex
  - Synexus Manchester Clinical Research Centre-Manchester Science Park, Manchester, Greater Manchester
  - Royal Oldham Hospital, Oldham, Greater Manchester
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - Lister Hospital, Stevenage, Hertfordshire
  - Queen Elizabeth II Hospital, East and North Hertfordshire NHS Trust, Welwyn Garden City, Hertfordshire
  - Medway Maritime Hospital, Gillingham, KENT
  - Synexus Scotland Clinical Research Centre, Glasgow, Lanarkshire
  - Bolton NHS Foundation Trust, Bolton, Lancashire
  - Synexus Lancashire Clinical Research Centre, Chorley, Lancashire
  - Layton Medical Centre, Layton, Blackpool, Lancashire
  - Synexus Merseyside Clinical Research Centre, Liverpool, Merseyside
  - Whitby Group Practice, Whitby, North Yorkshire
  - Albany House Medical Centre, Wellingborough, Northants
  - Southern Health & Social Care Trust, Craigavon Area Hospital, Portadown, Northern Ireland
  - Synexus North East Clinical Research Centre - Hexham General Hospital, Hexham, Northumberland
  - South Axholme Practice, Doncaster, South Yorkshire
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester, South Yorkshire
  - The Crouch Oak Family Practice, Addlestone, Surrey
  - Ely Bridge Surgery, Cardiff, Wales
  - Synexus Midlands Clinical Research Centre, Birmingham, WEST Midlands
  - City Hospital, Birmingham, WEST Midlands
  - Prince Philip Hospital, Llanelli, WEST Wales
  - Royal Free London NHS Foundation Trust, Barnet
  - Laurie Pike Health Centre, Birmingham
  - Heart of England NHS Foundation Trust, Dept. of Clinical Biochemistry & Immunology, Birmingham
  - Synexus Wales Clinical Research Centre, Cardiff
  - Ashgate Medical Practice, Chesterfield
  - Little Common Surgery, East Sussex
  - Sea Road Surgery, East Sussex
  - Staploe Medical Centre, Ely
  - McGlone Practice - Ballieston Health Centre, Glasgow
  - The Queen Elizabeth University Hospital- NHS Greater Glasgow and Clyde, Glosgow
  - Burbage Surgery, Hinckley
  - The Royal Liverpool and Broadgreen -University Hospitals NHS, Liverpool
  - Barts Health NHS Trust, London
  - Royal Free Hospital, London
  - Peart-Rose Research Unit, Hammersmith Hospital, Imperial College NHS Trust, London
  - The Red Porto cabin, The James Cook University Hospital, Middlesbrough
  - St Mary's Hospital, Newport
  - Wansford And Kings Cliffe Practice, Peterborough
  - Rothwell and Desborough Healthcare Group, Rothwell, Northants
  - Abertawe Bro Morgannwg University Local Health Board Joint, Swansea
  - Western Sussex Hosptials NHS Trust, Worthing
  - York Medical Group, York
  - Strensall Healthcare Centre, York

REFERENCES:
- [Derived] Chasman DI, Hyde CL, Giulianini F, Danning RD, Wang EQ, Hickling T, Ridker PM, Loomis AK. Genome-wide pharmacogenetics of anti-drug antibody response to bococizumab highlights key residues in HLA DRB1 and DQB1. Sci Rep. 2022 Mar 11;12(1):4266. doi: 10.1038/s41598-022-07997-5. PMID 35277540
- [Derived] Pradhan AD, Aday AW, Rose LM, Ridker PM. Residual Inflammatory Risk on Treatment With PCSK9 Inhibition and Statin Therapy. Circulation. 2018 Jul 10;138(2):141-149. doi: 10.1161/CIRCULATIONAHA.118.034645. Epub 2018 May 1. PMID 29716940
- [Derived] Ridker PM, Rose LM, Kastelein JJP, Santos RD, Wei C, Revkin J, Yunis C, Tardif JC, Shear CL; Studies of PCSK9 Inhibition and the Reduction of vascular Events (SPIRE) Investigators. Cardiovascular event reduction with PCSK9 inhibition among 1578 patients with familial hypercholesterolemia: Results from the SPIRE randomized trials of bococizumab. J Clin Lipidol. 2018 Jul-Aug;12(4):958-965. doi: 10.1016/j.jacl.2018.03.088. Epub 2018 Apr 3. PMID 29685591
- [Derived] Ridker PM, Revkin J, Amarenco P, Brunell R, Curto M, Civeira F, Flather M, Glynn RJ, Gregoire J, Jukema JW, Karpov Y, Kastelein JJP, Koenig W, Lorenzatti A, Manga P, Masiukiewicz U, Miller M, Mosterd A, Murin J, Nicolau JC, Nissen S, Ponikowski P, Santos RD, Schwartz PF, Soran H, White H, Wright RS, Vrablik M, Yunis C, Shear CL, Tardif JC; SPIRE Cardiovascular Outcome Investigators. Cardiovascular Efficacy and Safety of Bococizumab in High-Risk Patients. N Engl J Med. 2017 Apr 20;376(16):1527-1539. doi: 10.1056/NEJMoa1701488. Epub 2017 Mar 17. PMID 28304242
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481038&StudyName=The%20Evaluation%20Of%20PF-04950615%20%28RN316%29%20In%20Reducing%20The%20Occurrence%20Of%20Major%20Cardiovascular%20Events%20In%20High%20Risk%20Subjects

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial was terminated prematurely on November 1, 2016, due to the emerging clinical profile and the evolving treatment and market landscape for lipid-lowering agents.
Groups:
- Placebo: Participants received single dose of placebo matched to PF-04950615 subcutaneous injection once in every 2 weeks over a period of 3 years. Participants were followed up to 40 days after the last dose.
- Bococizumab (PF-04950615): Participants received single dose of PF-04950615, 150 milligrams, subcutaneous injection once in every 2 weeks over a period of 3 years. Participants were followed up to 40 days after the last dose.
Period: Overall Study
Arm/Group | Placebo | Bococizumab (PF-04950615)
Started | 5283 | 5281
Treated | 5279 | 5276
Completed | 5031 | 5045
Not Completed | 252 | 236
Not completed — Adverse Event | 10 | 6
Not completed — Death | 61 | 54
Not completed — Lost to Follow-up | 81 | 86
Not completed — Withdrawal by Subject | 90 | 76
Not completed — Other | 6 | 9
Not completed — Randomized, not treated | 4 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all participants who were randomized, excluding who attempted to be randomized more than once into a bococizumab cardiovascular (CV) outcomes trial (B1481022/B1481038) or attempted to be randomized in more than 1 CV outcomes trial and all participants enrolled at study Site 3027 where a quality-related event was identified.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bococizumab (PF-04950615) | Total
Number analyzed (Participants) | 5283 | 5281 | 10564
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (9.5) | 62.2 (9.6) | 62.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1849 | 1792 | 3641
  Male | 3434 | 3489 | 6923
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full analysis set (FAS): all participants who were randomized, excluding who attempted to be randomized more than once into a bococizumab cardiovascular (CV) outcomes trial (B1481022/B1481038) or attempted to be randomized in more than 1 CV outcomes trial and all participants enrolled at study Site 3027 where a quality-related event was identified.
  Participants
    Hispanic or Latino | 852 | 892 | 1744
    Not Hispanic or Latino | 4430 | 4387 | 8817
    Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: FAS: all participants who were randomized, excluding who attempted to be randomized more than once into a bococizumab cardiovascular (CV) outcomes trial (B1481022/B1481038) or attempted to be randomized in more than 1 CV outcomes trial and all participants enrolled at study Site 3027 where a quality-related event was identified.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 118 | 105 | 223
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 246 | 252 | 498
    White | 4776 | 4784 | 9560
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 143 | 140 | 283

OUTCOME MEASURES:

1. Primary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Major Cardiovascular (CV) Event
Description: Event rate per 100 participant-years for first occurrence of major CV event (adjudicated by Adjudication Committee) was reported. Major CV event was defined as any of the following: CV death [defined as sudden cardiac death, fatal myocardial infarction (MI), death due to heart failure, death due to stroke (fatal ischemic stroke or fatal stroke of undetermined etiology), or death due to other CV causes] non-fatal MI, non-fatal stroke, and hospitalization for unstable angina needing urgent revascularization. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of major CV event (maximum duration: up to 3.4 years)
Population: FAS: all participants who were randomized, excluding who attempted to be randomized more than once into a bococizumab CV outcomes trial (B1481022/B1481038) or attempted to be randomized in more than 1 CV outcomes trial and all participants enrolled at study Site 3027 where a quality-related event was identified.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 4.19 [3.66 to 4.78] | 3.33 [2.86 to 3.86]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Hazard ratio and 95% Confidence Interval (CI) were obtained from a Cox proportional hazards model stratified by geographic region and complete statin intolerance with treatment as a covariate; Test type: Superiority; p = 0.021469, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.97]

2. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Composite Endpoint of Cardiovascular (CV) Death, Non-fatal Myocardial Infraction (MI) or Non-fatal Stroke
Description: Event rate per 100 participant-years for first occurrence of composite endpoint of CV Death, non-fatal MI or non-fatal stroke (adjudicated by Adjudication Committee) was reported. CV death was defined as sudden cardiac death, fatal MI, death due to heart failure, death due to stroke (fatal ischemic stroke or fatal stroke of undetermined etiology), or death due to other CV causes. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of CV death, non-fatal MI or non-fatal stroke (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 3.58 [3.09 to 4.12] | 2.67 [2.25 to 3.14]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Hazard ratio and 95% CI were obtained from a Cox proportional hazards model stratified by geographic region and complete statin intolerance with treatment as a covariate; Test type: Superiority; p = 0.007597, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.60 to 0.93]

3. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Composite Endpoint of All-cause Death, Non-fatal Myocardial Infraction (MI), Non-fatal Stroke or Hospitalization for Unstable Angina Needing Urgent Revascularization
Description: Event rate per 100 participant-years for first occurrence of composite endpoint of all-cause death, non-fatal MI, non-fatal stroke or hospitalization for unstable angina needing urgent revascularization (adjudicated by Adjudication Committee) was reported. All-cause death was defined as the death due to any cause during the course of study. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of all-cause death, non-fatal MI, non-fatal stroke or hospitalization for unstable angina needing urgent revascularization (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 4.59 [4.03 to 5.20] | 3.76 [3.26 to 4.32]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.035958, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.68 to 0.99]

4. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Composite Endpoint of All-cause Death, Non-fatal Myocardial Infarction (MI) or Non-fatal Stroke
Description: Event rate per 100 participant-years for first occurrence of composite endpoint of all-cause death, non-fatal MI or non-fatal stroke (adjudicated by Adjudication Committee) was reported. All-cause death was defined as the death due to any cause during the course of study. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of all-cause death, non-fatal MI or non-fatal stroke (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 3.97 [3.45 to 4.54] | 3.09 [2.64 to 3.60]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.015694, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.64 to 0.95]

5. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Hospitalization for Unstable Angina Needing Urgent Revascularization
Description: Event rate per 100 participant-years for first occurrence of hospitalization for unstable angina needing urgent revascularization (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of hospitalization for unstable angina needing urgent revascularization (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.77 [0.56 to 1.05] | 0.73 [0.52 to 1.00]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.814224, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.62 to 1.46]

6. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Composite Endpoint of Cardiovascular (CV) Death, Non-fatal Myocardial Infarction (MI), Non-fatal Stroke or Hospitalization for Unstable Angina
Description: Event rate per 100 participant-years for first occurrence of composite endpoint of CV death, non-fatal MI, non-fatal stroke or hospitalization for unstable angina (adjudicated by Adjudication Committee) was reported. CV death was defined as sudden cardiac death, fatal MI, death due to heart failure, death due to stroke (fatal ischemic stroke or fatal stroke of undetermined etiology), or death due to other CV causes. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of CV death, non-fatal MI, non-fatal stroke or hospitalization for unstable angina (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 4.35 [3.81 to 4.94] | 3.45 [2.97 to 3.98]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.018053, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.96]

7. Secondary Outcome: Event Rate Per 100 Participant-years for Cardiovascular (CV) Death
Description: Event rate per 100 participant-years for occurrence of CV death (adjudicated by Adjudication Committee) was reported. CV death was defined as sudden cardiac death, fatal MI, death due to heart failure, death due to stroke (fatal ischemic stroke or fatal stroke of undetermined etiology), or death due to other CV causes. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of adjudicated and confirmed occurrence of CV death (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.62 [0.43 to 0.87] | 0.51 [0.34 to 0.74]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.446033, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.50 to 1.36]

8. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Any Myocardial Infarction (Fatal or Non-fatal)
Description: Event rate per 100 participant-years for first occurrence of any myocardial infarction (fatal or non-fatal) (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of any myocardial infarction (fatal or non-fatal) (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 2.39 [2.00 to 2.84] | 1.79 [1.45 to 2.19]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.029977, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.57 to 0.97]

9. Secondary Outcome: Event Rate Per 100 Participant-years for Fatal Myocardial Infarction (MI)
Description: Event rate per 100 participant-years for occurrence of fatal MI (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of adjudicated and confirmed occurrence of fatal MI (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.16 [0.08 to 0.31] | 0.07 [0.02 to 0.19]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.162615, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.14 to 1.44]

10. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Non-fatal Myocardial Infarction (MI)
Description: Event rate per 100 participant-years for first occurrence of non-fatal MI (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of non-fatal MI (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 2.26 [1.88 to 2.70] | 1.74 [1.40 to 2.12]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.051534, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.59 to 1.00]

11. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Any Stroke (Fatal or Non-fatal)
Description: Event rate per 100 participant-years for first occurrence of any stroke (fatal or non-fatal) (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of any stroke (fatal or non-fatal) (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.72 [0.51 to 0.98] | 0.48 [0.31 to 0.70]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.104998, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.41 to 1.09]

12. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Any Stroke (Fatal or Non-fatal), of Any Etiology
Description: Event rate per 100 participant-years for first occurrence of any stroke (fatal or non-fatal) of any etiology (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of any stroke (fatal or non-fatal) of any etiology (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.77 [0.56 to 1.04] | 0.61 [0.42 to 0.85]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.294331, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.50 to 1.24]

13. Secondary Outcome: Event Rate Per 100 Participant-years for Fatal Stroke
Description: Event rate per 100 participant-years for occurrence of fatal stroke (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of adjudicated and confirmed occurrence of fatal stroke (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.00 [0.00 to 0.05] | 0.00 [0.00 to 0.05]

14. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Non-fatal Stroke
Description: Event rate per 100 participant-years for first occurrence of non-fatal stroke (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of non-fatal stroke (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.72 [0.51 to 0.98] | 0.48 [0.31 to 0.70]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.104998, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.41 to 1.09]

15. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Hospitalization for Unstable Angina
Description: Event rate per 100 participant-years for first occurrence of hospitalization for unstable angina (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of hospitalization for unstable angina (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.94 [0.70 to 1.24] | 0.85 [0.62 to 1.13]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.601200, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.60 to 1.34]

16. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Hospitalization for Congestive Heart Failure (CHF)
Description: Event rate per 100 participant-years for first occurrence of hospitalization for CHF (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of hospitalization for CHF (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.75 [0.54 to 1.02] | 0.83 [0.60 to 1.11]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.678061, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.72 to 1.67]

17. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Coronary Revascularization
Description: Event rate per 100 participant-years for first occurrence of coronary revascularization (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of coronary revascularization (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 4.18 [3.65 to 4.77] | 3.23 [2.76 to 3.75]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.010457, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.63 to 0.94]

18. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Coronary Artery Bypass Graft Surgery (CABG)
Description: Event rate per 100 participant-years for first occurrence of CABG (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of CABG (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 0.48 [0.31 to 0.70] | 0.57 [0.39 to 0.81]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.509847, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.71 to 2.01]

19. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Percutaneous Coronary Intervention (PCI)
Description: Event rate per 100 participant-years for first occurrence of PCI (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of PCI (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 3.73 [3.23 to 4.28] | 2.70 [2.27 to 3.17]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.002981, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.90]

20. Secondary Outcome: Event Rate Per 100 Participant-years for First Occurrence of Any Arterial Revascularizations
Description: Event rate per 100 participant-years for first occurrence of any arterial revascularizations (adjudicated by Adjudication Committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of any arterial revascularizations (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 1.51 [1.20 to 1.88] | 1.44 [1.14 to 1.80]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.748975, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.70 to 1.30]

21. Secondary Outcome: Event Rate Per 100 Participant-years for All-cause Death
Description: Event rate per 100 participant-years for occurrence of all-cause death (adjudicated by Adjudication Committee) was reported. All-cause death was defined as the death due to any cause during the course of study. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of adjudicated and confirmed occurrence of all-cause death (maximum duration: up to 3.4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 participant-years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Events per 100 participant-years | 1.06 [0.81 to 1.37] | 0.97 [0.73 to 1.27]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.626157, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.63 to 1.32]

22. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 14
Time Frame: Baseline, Week 14
Population: Analysis was performed on FAS. Here, "Number of participants analyzed" (N) signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 4712 | 4654
Percent change | 2.13 (0.36) | -54.77 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Least square (LS) mean differences, associated 95% CI, and p-values were from an mixed model repeated measures (MMRM) model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, MMRM; LS mean difference = -56.90, 95% CI 2-sided [-57.91 to -55.89], Standard Error of Mean 0.51

23. Secondary Outcome: Nominal Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 14
Time Frame: Baseline, Week 14
Population: Analysis was performed on FAS. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 4712 | 4654
mg/dL | 0.69 (0.47) | -73.11 (0.47)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); LS mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, MMRM; LS mean difference = -73.80, 95% CI 2-sided [-75.11 to -72.50], Standard Error of Mean 0.67

24. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Last Post-baseline Measurement
Time Frame: Baseline, last post-baseline measurement (any time up to Week 140)
Population: Analysis was performed on FAS. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5242 | 5246
Percent change | 2.90 (0.45) | -36.41 (0.45)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); LS-mean difference, associated 95% CI, and p-value were from an analysis of covariance (ANCOVA) model with fixed effects for treatment group, baseline value, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = -39.31, 95% CI 2-sided [-40.55 to -38.06], Standard Error of Mean 0.64

25. Secondary Outcome: Percent Change From Baseline in Lipid Levels at Week 14
Description: Lipids included non-high density lipoprotein cholesterol (non-HDL-C), very low density lipoprotein cholesterol (VLDL-C), remnant lipoprotein cholesterol (RLP-C), apolipoprotein B (Apo B), HDL-C, apolipoprotein A-I (Apo A-I) and total cholesterol.
Time Frame: Baseline, Week 14
Population: FAS population. Here, number analyzed "n" signifies number of participants who were evaluable for the specified categories.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Percent change
  Non-HDL-C: number analyzed (Participants) | 4698 | 4646
  Non-HDL-C | 1.82 (0.34) | -50.05 (0.34)
  VLDL-C: number analyzed (Participants) | 4711 | 4657
  VLDL-C | 4.88 (0.56) | -13.54 (0.56)
  RLP-C: number analyzed (Participants) | 4696 | 4635
  RLP-C | 8.76 (0.81) | -20.44 (0.81)
  Apo B: number analyzed (Participants) | 4616 | 4588
  Apo B | 1.89 (0.35) | -49.51 (0.35)
  HDL-C: number analyzed (Participants) | 4698 | 4647
  HDL-C | 1.05 (0.21) | 7.96 (0.21)
  Apo A-I: number analyzed (Participants) | 4617 | 4588
  Apo A-I | 0.07 (0.18) | 4.46 (0.18)
  Total cholesterol: number analyzed (Participants) | 4711 | 4658
  Total cholesterol | 1.26 (0.28) | -36.72 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Non-HDLC: LS-mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, MMRM; LS mean difference = -51.87, 95% CI 2-sided [-52.81 to -50.94], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: Placebo vs Bococizumab (PF-04950615); VLDL-C: LS-mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, MMRM; LS mean difference = -18.41, 95% CI 2-sided [-19.96 to -16.86], Standard Error of Mean 0.79
Statistical Analysis 3: Comparison: Placebo vs Bococizumab (PF-04950615); RLP-C: LS-mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, MMRM; LS mean difference = -29.20, 95% CI 2-sided [-31.44 to -26.96], Standard Error of Mean 1.14
Statistical Analysis 4: Comparison: Placebo vs Bococizumab (PF-04950615); Apo B: LS-mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 52 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, MMRM; LS mean difference = -51.40, 95% CI 2-sided [-52.37 to -50.42], Standard Error of Mean 0.50
Statistical Analysis 5: Comparison: Placebo vs Bococizumab (PF-04950615); HDL-C: LS-mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, MMRM; LS mean difference = 6.91, 95% CI 2-sided [6.33 to 7.50], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Placebo vs Bococizumab (PF-04950615); Apo A-I: LS-mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 52 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, MMRM; LS mean difference = 4.40, 95% CI 2-sided [3.90 to 4.90], Standard Error of Mean 0.25
Statistical Analysis 7: Comparison: Placebo vs Bococizumab (PF-04950615); Total cholesterol: LS-mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and complete statin intolerance; Test type: Superiority; p < 0.001, MMRM; LS mean difference = -37.99, 95% CI 2-sided [-38.75 to -37.22], Standard Error of Mean 0.39

26. Secondary Outcome: Percent Change From Baseline in Log-transformed Triglycerides and Lipoprotein (a) (Lp[a]) at Week 14
Time Frame: Baseline, Week 14
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5283 | 5281
Percent change
  Triglycerides: number analyzed (Participants) | 4711 | 4657
  Triglycerides | -1.4 (34.55) | -19.7 (30.71)
  Lp(a): number analyzed (Participants) | 4650 | 4598
  Lp(a) | -2.0 (31.03) | -33.3 (31.21)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Triglycerides: LS-mean differences, associated 95% CI and p-values were from an MMRM model including observations through Week 70 on the difference of log-transformed observations with fixed effects for treatment group, visit, treatment group*visit interaction, log-transformed baseline value, log-transformed baseline value*visit interaction, geographical region and complete statin intolerance. The 95% CI was derived by exponentiating the LS-mean difference confidence interval from the log scale; Test type: Superiority; p < 0.001, MMRM; LS mean difference = 0.82, 95% CI 2-sided [0.81 to 0.83]
Statistical Analysis 2: Comparison: Placebo vs Bococizumab (PF-04950615); Lp(a): LS-mean differences, associated 95% CI and p-values were from an MMRM model on the Difference of log-transformed observations with fixed effects for treatment group, visit, a treatment group*visit interaction, log-transformed baseline value, log-transformed baseline value*visit interaction, geographical region and complete statin intolerance. The 95% CI was derived by exponentiating the LS-mean difference confidence interval from the log scale; Test type: Superiority; p < 0.001, MMRM; LS mean difference = 0.68, 95% CI 2-sided [0.67 to 0.69]

27. Secondary Outcome: Percent Change From Baseline in Log-transformed High Sensitivity C-Reactive Protein (Hs-CRP) at Week 14
Time Frame: Baseline, Week 14
Population: Analysis was performed on FAS. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 4655 | 4620
Percent change | -4.8 (83.68) | 0.3 (90.03)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); LS-mean differences, associated 95% CI and p-values were from an MMRM model on the difference of log-transformed observations with fixed effects for treatment group, visit, treatment group*visit interaction, log-transformed baseline value, log-transformed baseline value*visit interaction, geographical region and complete statin intolerance; Test type: Superiority; p = 0.002, MMRM; LS mean difference = 1.06, 95% CI 2-sided [1.02 to 1.09]

ADVERSE EVENTS:
Time Frame: Baseline up to 3.4 years
Description: Safety analysis set: all participants who randomized, had atleast 1 dose of study drug, excluding those attempted to randomize more than once in a bococizumab CV outcomes trial (B1481022/B1481038) or attempted to randomize in more than 1 CV outcomes trial, and all participants enrolled at study Site 3027 where a quality-related event was identified
Arm/Group | Placebo | Bococizumab (PF-04950615)
All-Cause Mortality (participants affected / at risk) | 61/5279 | 54/5276
Serious Adverse Events (participants affected / at risk) | 994/5279 | 934/5276
Other Adverse Events (participants affected / at risk) | 2128/5279 | 2453/5276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=5279) | Bococizumab (PF-04950615) (N=5276)
Anaemia (Blood and lymphatic system disorders) | 4 | 6
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 3
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 7 | 9
Acute left ventricular failure (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 40 | 30
Angina pectoris (Cardiac disorders) | 92 | 64
Angina unstable (Cardiac disorders) | 93 | 73
Anginal equivalent (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 3 | 3
Arrhythmia (Cardiac disorders) | 3 | 4
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 3
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 34 | 26
Atrial flutter (Cardiac disorders) | 9 | 5
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 3 | 4
Atrioventricular block complete (Cardiac disorders) | 1 | 4
Atrioventricular block second degree (Cardiac disorders) | 3 | 1
Bradycardia (Cardiac disorders) | 7 | 1
Cardiac arrest (Cardiac disorders) | 5 | 4
Cardiac failure (Cardiac disorders) | 15 | 16
Cardiac failure acute (Cardiac disorders) | 0 | 3
Cardiac failure chronic (Cardiac disorders) | 3 | 2
Cardiac failure congestive (Cardiac disorders) | 31 | 24
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 31 | 29
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 5 | 5
Coronary artery stenosis (Cardiac disorders) | 17 | 7
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Dressler's syndrome (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 2 | 0
Left ventricular failure (Cardiac disorders) | 3 | 1
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 52 | 34
Myocardial ischaemia (Cardiac disorders) | 10 | 9
Palpitations (Cardiac disorders) | 2 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 4 | 4
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 3
Systolic dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 3 | 6
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 5 | 5
Hydrocele (Congenital, familial and genetic disorders) | 0/3434 | 1/3489 — This event was gender specific.
Phimosis (Congenital, familial and genetic disorders) | 1/3434 | 0/3489 — This event was gender specific.
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 3
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 1
Addison's disease (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Thyroid mass (Endocrine disorders) | 0 | 2
Amaurosis fugax (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 2
Diabetic retinopathy (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Macular fibrosis (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 1 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0
Retinal infarction (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 1
Coeliac artery stenosis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Diverticulum oesophageal (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 2
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 5 | 5
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1/1849 | 0/1792 — This event was gender specific.
Inguinal hernia (Gastrointestinal disorders) | 2 | 4
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 1
Lip disorder (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 4
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 4 | 6
Pancreatitis acute (Gastrointestinal disorders) | 4 | 3
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Reactive gastropathy (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 3
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 5
Strangulated umbilical hernia (Gastrointestinal disorders) | 0/1849 | 1/1792 — This event was gender specific.
Ulcerative gastritis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 2/1849 | 1/1792 — This event was gender specific.
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0/1849 | 1/1792 — This event was gender specific.
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 4
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 3 | 1
Cardiac death (General disorders) | 1 | 0
Chest discomfort (General disorders) | 3 | 1
Chest pain (General disorders) | 14 | 8
Complication associated with device (General disorders) | 1 | 1
Death (General disorders) | 6 | 9
Drug withdrawal syndrome (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Ill-defined disorder (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 1
Inflammation (General disorders) | 1 | 0
Multi-organ disorder (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 50 | 32
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 2 | 0
Peripheral swelling (General disorders) | 2 | 0
Polyp (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Stenosis (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 8 | 5
Sudden death (General disorders) | 3 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Vascular stent restenosis (General disorders) | 2 | 1
Vascular stent stenosis (General disorders) | 1 | 2
Vascular stent thrombosis (General disorders) | 0 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Biliary fistula (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 6 | 5
Cholecystitis acute (Hepatobiliary disorders) | 4 | 4
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 7 | 5
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Immunosuppression (Immune system disorders) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 1 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 2
Anal abscess (Infections and infestations) | 0 | 4
Appendicitis (Infections and infestations) | 5 | 4
Arteriovenous graft site infection (Infections and infestations) | 2 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 0
Bacterial diarrhoea (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 7 | 5
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Cardiac valve vegetation (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 10 | 8
Cholecystitis infective (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 2
Clostridium difficile infection (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 0 | 2
Device related infection (Infections and infestations) | 0 | 2
Diabetic foot infection (Infections and infestations) | 2 | 2
Diabetic gangrene (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 5 | 6
Endocarditis (Infections and infestations) | 2 | 2
Epididymitis (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 2 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastritis viral (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 6 | 2
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 3
Groin abscess (Infections and infestations) | 1 | 1
Groin infection (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 1
Hepatic cyst infection (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Incision site infection (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 3
Infectious colitis (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 4
Lower respiratory tract infection (Infections and infestations) | 4 | 1
Lung abscess (Infections and infestations) | 1 | 0
Medical device site abscess (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 3 | 4
Otitis externa (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 35 | 28
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0
Post procedural pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelocystitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 5
Pyelonephritis acute (Infections and infestations) | 0 | 2
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2
Scrotal abscess (Infections and infestations) | 1 | 1
Sebaceous gland infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 13
Septic shock (Infections and infestations) | 3 | 2
Sinusitis (Infections and infestations) | 1 | 2
Sinusitis bacterial (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tick-borne viral encephalitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 15 | 9
Urosepsis (Infections and infestations) | 1 | 3
Viral infection (Infections and infestations) | 1 | 0
Viral sepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 2 | 2
Acoustic shock (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Dural tear (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 5
Femur fracture (Injury, poisoning and procedural complications) | 5 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 3 | 2
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Gallbladder injury (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 4 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 2
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Suture related complication (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 2
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 2
Wound (Injury, poisoning and procedural complications) | 2 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 2 | 1
Blood ketone body increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 2 | 0
Ejection fraction abnormal (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Exercise test abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 2
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 2 | 1
Myocardial necrosis marker increased (Investigations) | 0 | 1
Neurological examination (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0
Renal function test abnormal (Investigations) | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 1
Stress echocardiogram abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 5
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 3
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8 | 7
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 | 17
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Peripheral arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 | 1
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 3
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/1849 | 2/1792 — This event was gender specific.
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1849 | 0/1792 — This event was gender specific.
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3434 | 1/3489 — This event was gender specific.
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13/3434 | 11/3489 — This event was gender specific.
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1849 | 1/1792 — This event was gender specific.
Amputation stump pain (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Basal ganglia stroke (Nervous system disorders) | 0 | 1
Brain stem haemorrhage (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 14 | 12
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 2 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 10 | 7
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 6 | 3
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Fahr's disease (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 3
Haemorrhagic stroke (Nervous system disorders) | 2 | 5
Headache (Nervous system disorders) | 2 | 4
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegic migraine (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 3 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 2
Ischaemic neuropathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 23 | 16
Lacunar infarction (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 1 | 1
Monoplegia (Nervous system disorders) | 0 | 1
Nerve root compression (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Neuritis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 3
Radicular syndrome (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 2 | 3
Seizure (Nervous system disorders) | 2 | 2
Sensory disturbance (Nervous system disorders) | 0 | 2
Serotonin syndrome (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 1
Subarachnoid haematoma (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 16 | 18
Thrombotic stroke (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 16 | 14
Vertebral artery stenosis (Nervous system disorders) | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0/1849 | 1/1792 — This event was gender specific.
Device dislocation (Product Issues) | 1 | 1
Device malfunction (Product Issues) | 1 | 0
Device material issue (Product Issues) | 0 | 1
Manufacturing issue (Product Issues) | 0 | 1
Thrombosis in device (Product Issues) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 2
Alcoholism (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Delirium tremens (Psychiatric disorders) | 0 | 1
Delusional disorder, unspecified type (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 4 | 6
Drug abuse (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 2
Neurologic somatic symptom disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 3
Suicide attempt (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 15 | 10
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Bladder diverticulum (Renal and urinary disorders) | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 6 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal artery thrombosis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 2 | 2
Renal failure (Renal and urinary disorders) | 3 | 3
Renal impairment (Renal and urinary disorders) | 0 | 2
Stress urinary incontinence (Renal and urinary disorders) | 1 | 1
Ureterolithiasis (Renal and urinary disorders) | 3 | 2
Urethral disorder (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 4 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/3434 | 2/3489 — This event was gender specific.
Breast hyperplasia (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1/1849 | 0/1792 — This event was gender specific.
Cystocele (Reproductive system and breast disorders) | 0/1849 | 1/1792 — This event was gender specific.
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0/1849 | 1/1792 — This event was gender specific.
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/1849 | 1/1792 — This event was gender specific.
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1/1849 | 0/1792 — This event was gender specific.
Prostatitis (Reproductive system and breast disorders) | 5/3434 | 2/3489 — This event was gender specific.
Rectocele (Reproductive system and breast disorders) | 1/1849 | 1/1792 — This event was gender specific.
Uterine haemorrhage (Reproductive system and breast disorders) | 0/1849 | 1/1792 — This event was gender specific.
Uterine prolapse (Reproductive system and breast disorders) | 0/1849 | 1/1792 — This event was gender specific.
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 3
Idiopathic angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Peau d'orange (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 2
Immobile (Social circumstances) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 4
Aortic occlusion (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 8 | 4
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0
Arterial rupture (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 2 | 0
Arteriosclerosis (Vascular disorders) | 1 | 2
Axillary vein thrombosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 2
Diabetic vascular disorder (Vascular disorders) | 1 | 0
Dry gangrene (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 1 | 0
Femoral artery embolism (Vascular disorders) | 1 | 0
Granulomatosis with polyangiitis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 4 | 2
Hypertension (Vascular disorders) | 6 | 4
Hypertensive crisis (Vascular disorders) | 5 | 7
Hypertensive emergency (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 5 | 7
Iliac artery occlusion (Vascular disorders) | 0 | 2
Infarction (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 4 | 3
Internal haemorrhage (Vascular disorders) | 1 | 0
Labile hypertension (Vascular disorders) | 1 | 0
Microangiopathy (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 13 | 14
Peripheral artery occlusion (Vascular disorders) | 6 | 1
Peripheral artery stenosis (Vascular disorders) | 3 | 8
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 8 | 4
Peripheral vascular disorder (Vascular disorders) | 14 | 10
Shock (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 1 | 1
Vascular pain (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5279) | Bococizumab (PF-04950615) (N=5276)
Injection site reaction (General disorders) | 68 | 617
Angina pectoris (Cardiac disorders) | 120 | 104
Diarrhoea (Gastrointestinal disorders) | 136 | 133
Fatigue (General disorders) | 134 | 141
Injection site erythema (General disorders) | 23 | 164
Non-cardiac chest pain (General disorders) | 111 | 89
Bronchitis (Infections and infestations) | 159 | 167
Influenza (Infections and infestations) | 112 | 157
Nasopharyngitis (Infections and infestations) | 227 | 236
Upper respiratory tract infection (Infections and infestations) | 170 | 180
Urinary tract infection (Infections and infestations) | 107 | 137
Fall (Injury, poisoning and procedural complications) | 156 | 141
Diabetes mellitus (Metabolism and nutrition disorders) | 167 | 147
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 126 | 109
Arthralgia (Musculoskeletal and connective tissue disorders) | 182 | 211
Back pain (Musculoskeletal and connective tissue disorders) | 180 | 182
Muscle spasms (Musculoskeletal and connective tissue disorders) | 109 | 108
Myalgia (Musculoskeletal and connective tissue disorders) | 208 | 233
Pain in extremity (Musculoskeletal and connective tissue disorders) | 120 | 125
Dizziness (Nervous system disorders) | 143 | 136
Headache (Nervous system disorders) | 163 | 171
Cough (Respiratory, thoracic and mediastinal disorders) | 104 | 118
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 124 | 96
Hypertension (Vascular disorders) | 242 | 226

LIMITATIONS AND CAVEATS:
As specified in statistical analysis plan, due to discontinuation of the bococizumab clinical development program, health care resource utilization endpoints were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT01975389/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT01975389/SAP_001.pdf